## Mayo Clinic Cancer Center

# MC1941 - Phase II Trial of Trifluridine/Tipiracil in Combination with Irinotecan in Biliary Tract Cancers

Sponsor/Principal Investigator: Amit Mahipal MBBS

Co-Investigators:

Statistician:

FDA IND #: EXEMPT (144800)

## **Trial Supported by:**

Funding: NCCN Oncology Research Program through a research grant provided by Taiho Oncology, Inc.

## **Drug Availability:**

**Supplied Investigational Agents:** trifluridine/tipiracil (TAS-102; Lonsurf®)

Commercial Agents: irinotecan

Document History<br/>Activation(Effective Date)MCCC Amendment 118Oct201918May2020

√Study contributor(s) not responsible for patient care

Protocol Version Date: 14Apr2020

# **Protocol Resources**

| Questions: | Contact 1 | Name: |
|---|---|---|
| Patient eligibility*, test schedule, treatment delays/ interruptions/ adjustments, dose modifications, adverse events, forms completion and submission | | |
| Drug administration, infusion pumps, nursing guidelines | | |
| Clinical and Data Coordinators | Data Coordinators | Clinical Coordinators |
| Protocol document, consent form, regulatory issues | | |
| Laboratory | TBD Laboratory Contact for Correlative S Phone: 507/ Email: | Studies |
| Serious Adverse Event Reporting | | |

<sup>\*</sup>No waivers of eligibility allowed

# **Table of Contents**

| | 1 - Phase II Trial of Trifluridine/Tipiracil in Combination with Irinotecan in Bi | |
|---|---|---|
| | Resources | |
| | Contents | |
| 1.0 | Background | |
| 2.0 | Goals | |
| 3.0 | Registration Patient Eligibility | |
| 4.0 | Test Schedule | 11 |
| 5.0 | Stratification Factors OR Grouping Factor: None | 12 |
| 6.0 | Registration Procedures | |
| 7.0 | Protocol Treatment | 14 |
| 8.0 | Dosage Modification Based on Adverse Events | 16 |
| 9.0 | Ancillary Treatment/Supportive Care | 19 |
| 10.0 | Adverse Event (AE) Monitoring and Reporting | 20 |
| 11.0 | Treatment Evaluation/Measurement of Effect | 34 |
| 12.0 | Descriptive Factors | 39 |
| 13.0 | Treatment/Follow-up Decision at Evaluation of Patient | 39 |
| 14.0 | Body Fluid Biospecimens | 41 |
| 15.0 | Drug Information | 45 |
| 16.0 | Statistical Considerations and Methodology | 51 |
| 17.0 | Pathology Considerations/Tissue Biospecimens | 57 |
| 18.0 | Records and Data Collection Procedures | 61 |
| 19.0 | Budget | 62 |
| 20.0 | References | 63 |
| Appendi | ix I ECOG Performance Status | 66 |
| Appendi | ix II Patient Medication Diary | 67 |

## Schema



Cycle = 14 days

Generic name: trifluridine/tipiracil (FTD/TPI; TAS-102)
Brand name(s): Lonsurf®
Mayo Abbreviation: FTD/TPI
Availability: Supplied by Taiho Pharmaceuticals

Generic name: irinotecan
Brand name(s): Camptosar®
Mayo Abbreviation:
Availability: Commercial

## 1.0 Background

## 1.1 Biliary Tract Cancer

Biliary tract cancers (BTCs) include malignant intrahepatic and extrahepatic cholangiocarcinomas, gallbladder and ampullary cancers. It is estimated that 12,190 patients will be diagnosed with BTCs in 2018 in United States. (Siegel et al. 2018) Most patients with BTCs present with unresectable or metastatic disease. Even in patients with resectable disease, the recurrences are frequent. The median survival of patients with advanced BTCs is less than 4.5 months. (Glimelius et al. 1996; Sharma et al. 2010) Combination gemcitabine and cisplatin has been established as first line standard of care treatment based on the Advanced Biliary Tract Cancer-02 (ABC-02) phase III trial. (Valle et al. 2010) Unfortunately, the median overall survival (OS) was less than a year in this trial. There is no FDA-approved second line option for patients with advanced BTCs. There is a huge unmet need to develop novel therapies to improve outcome for patients diagnosed with BTCs.

## 1.2 Trifluridine/tipiracil

Trifluridine/tipiracil is a novel oral nucleoside consisting of  $\alpha$ ,  $\alpha$ ,  $\alpha$ -trifluorothymidine (trifluridine) and 5-chloro-6-(2-iminopyrrolidin-1-yl) methyl-2,4 (1H,3H)-pyrimidinedione hydrochloride (tipiracil). The active antitumor component is trifluridine which inhibits thymidylate synthase and is incorporated into DNA in tumor cells. Tipiracil is a thymidine phosphorylase inhibitor which prevents trifluridine from degradation. Therefore, trifluridine/tipiracil is mechanistically different from 5-fluorouracil (5-FU).

The clinical safety and efficacy of trifluridine/tipiracil was evaluated in the RECOURSE study conducted in patients with previously treated metastatic colorectal cancer (mCRC). (Mayer et al. 2015) A total of 800 patients were randomized to receive trifluridine/tipiracil plus best supportive care (BSC) or placebo plus BSC. Patients received 35 mg/m<sup>2</sup> trifluridine/tipiracil or matching placebo orally twice daily after meals on Days 1-5 and 8-12 of each 28-day cycle until disease progression or unacceptable toxicity. The RECOURSE study met the efficacy endpoints of significant improvement in OS and PFS compared to placebo in patients with refractory mCRC whose disease had progressed after standard therapies. The median OS was 7.1 months with trifluridine/tipiracil compared to 5.3 months in the placebo group (hazard ratio: 0.68; 95% CI: 0.56-0.78). Median PFS was 2 months in trifluridine/tipiracil group and 1.7 months in placebo group (hazard ratio: 0.48; 95% CI: 0.41-0.57). Common adverse events included fatigue, nausea, vomiting, diarrhea, anorexia and cytopenias. In addition, trifluridine/tipiracil also showed improved median OS compared to placebo in the phase 3 TAGS trial of 507 patients with refractory gastric and gastroesophageal junction cancer who had received at least two prior therapies. (Shitara et al. 2018)

The clinical activity of trifluridine/tipiracil has also been explored in combination with cytotoxic agents such as oxaliplatin and irinotecan in patients with mCRC whose disease progressed after at least one line of therapy. A phase I trial of trifluridine/tipiracil plus oxaliplatin in 17 patients with mCRC did not observe dose limiting toxicities (DLTs) with 23.5% Grade 3/4 neutropenia, 5.9% Grade 3/4, and 5.9% peripheral sensory neuropathy. These results were comparable to historical control. The recommended dose for phase II study was trifluridine/tipiracil 35 mg/m<sup>2</sup> BID (Days 1-5 every 2 weeks) with oxaliplatin 85 mg/m<sup>2</sup> (Day 1). Eight (47%) patients had stable disease. One (2.1%)

patient had a partial response. (Hollebecque et al. 2018) The combination of trifluridine/tipiracil and irinotecan was evaluated in 26 patients with advanced gastrointestinal tumors. The majority of patients had CRC (81%) whose disease progressed after at least one previous line of therapy. The study declared the maximum tolerated dose (MTD) as trifluridine/tipiracil 25 mg/m² on Days 1-5 and irinotecan 180 mg/m² on Day 1 every 14-day cycle based on two observed DLTs (Grade 3 fatigue and Grade 2 neutropenia) in the trifluridine/tipiracil 30 mg/m² and irinotecan 180 mg/m² cohort. In the subsequent dose expansion cohort of 24 patients with refractory mCRC treated with trifluridine/tipiracil, irinotecan, and bevacizumab, 10 (42%) patients had Grade 3/4 neutropenia, 3 (12.5%) patients had Grade 3/4 diarrhea. Three (12.5%) patients had a partial response and the disease control rate was 83% with median PFS of 7.9 months. (Varghese et al. 2018a; Varghese et al. 2018b)

## 1.3 Study Rationale

Fluoropyrimidine and irinotecan-based regimens are frequently utilized for treatment of advanced BTCs despite the fact that they are not FDA approved. (Huggett et al. 2014; Rogers et al. 2014) In retrospective studies, fluoropyrimidine based treatments have been shown to be associated with improved survival. (Huggett et al. 2014) However, there are only limited small prospective studies reported utilizing fluoropyrimidines. Single agent 5-FU in early trials has yielded response rates of 10% with median OS of approximately 6 months as a first line treatment. (Choi et al. 2000) S-1, a combination of tegafur (that is converted to 5-FU in the liver), 5-chloro-2,4-dihydroxypyridine (inhibitor of dihydropyrimidine dehydrogenase) and potassium oxonate has also shown modest activity in advanced BTCs as a single agent. (Ueno et al. 2004) The same applies to single agent irinotecan as demonstrated in a small phase 2 trial where the response rate of advanced BTCs was 8%. (Sanz-Altamira et al. 2001)

Combination therapies such as 5-FU or capecitabine plus irinotecan as 2<sup>nd</sup>-line therapy for advanced BCTs are associated with better response rates at the expense of increased toxicities. The combination of 5-FU and irinotecan in an early trial demonstrated a response rate of 10% in 17 patients. (Feisthammel et al. 2007) A more recent randomized phase 2 trial compared capecitabine plus irinotecan with irinotecan alone as 2<sup>nd</sup>-line therapy in 60 patients with advanced BTCs. The authors found that the capecitabine plus irinotecan arms showed a significantly higher response rate of 13.3% vs 6.7% and disease control rate of 63% vs 50% with a similar toxicity profile, other than hand-foot syndrome which is unique to capecitabine. (Zheng et al. 2018) Addition of other agents to this combination in the 2<sup>nd</sup>-line setting was proven to have non-superior activity but significantly increased toxicities. (Larsen et al. 2018; Guion-Dusserre et al. 2015) These studies suggest that there may be a role for fluoropyrimidines in combination with irinotecan in advanced BTCs.

The mechanism of trifluridine/tipiracil is distinct from fluoropyrimidine, which provided several advantages over 5-FU. Clinically with a twice daily dosing schedule of trifluridine/tipiracil, incorporation into DNA is the primary mechanism of action for antitumor effects instead of thymidine synthase inhibition when it was given with continuous infusion as 5-FU. Tipiracil is a potent inhibitor of thymidine phosphorylase, which is the enzyme that degrades trifluridine and helps maintain adequate plasma concentration needed for its activity. Thereby, the antitumor activity of trifluridine is more sustained compared to 5-FU, whose inhibition of thymidylate synthase rapidly disappears after rapid drug elimination. (Lenz et al. 2015; Tanaka et al. 2014) Trifluridine/tipiracil has shown activity in both fluoropyrimidine sensitive and resistant

MC1941 7 MCCC Amendment 1

tumors. (Emura et al. 2004a; Emura et al. 2004b) The primary mechanism of resistance to 5-FU seems to be the decrease in activity of orotate phosphoribosyl transferase resulting in decrease in cellular uptake of 5-FU in the RNA fraction. (Murakami et al. 2000) There is no change in thymidylate synthase level. Trifluridine has demonstrated activity in 5-FU resistant colorectal and gastric cancer cell lines, as activity of trifluridine/tipiracil is not dependent on orotate phosphoribosyltransferase. (Lenz et al. 2015) Autophagy has also shown to play a role in resistance to 5-FU but not to trifluridine. (Bijnsdorp et al. 2010) The potential superiority of trifluridine/tipiracil to 5-FU has also be implicated in a randomized phase 2 trial of trifluridine/tipiracil with bevacizumab versus capecitabine with bevacizumab as first-line therapy in patients with metastatic CRC who were not eligible for intensive therapy. The trifluridine/tipiracil plus bevacizumab arm had longer median OS of 18.0 months versus 16.1 months in the capecitabine plus bevacizumab arm with HR 0.56 (95% CI: 0.32-0.98). (Lesniewski-Kmak et al. 2018)

Our group (PI: Amit Mahipal) has recently completed accrual of 28 patients from October 2017 to August 2018 to a phase 2 trial evaluating the single-agent activity of trifluridine/tipiracil in metastatic refractory BTCs (NCT03278106). Eligible patients had at least one gemcitabine-based chemotherapy and were treated with trifluridine/tipiracil at the dose of 35 mg/m² bid, Days 1-5 and 8-12 of a 28–day cycle. All patients received at least one (1) cycle of trifluridine/tipiracil. Median number of cycles received was 3 (range 1-8). The most common Grade 3 or worse adverse events were neutrophil count decreased (44.4%), anemia (22.2%), alkaline phosphatase increased (22.2%), blood bilirubin increased (18.5%), and white blood cell decreased (18.5%), without any unexpected safety signals. Among 27 evaluable patients for response, the best response was stable disease in 13 (48%) patients. PFS rate at 16 weeks was 9/27 [33.3%; 95% confidence interval (CI): 16.5-54.0%]. Median PFS and OS were 3.9 (2.0-6.7) and 6.8 (5.8-12.3) months, respectively.

The early toxicities and efficacy data from our study on single-agent trifluridine/tipiracil in advanced BTCs and previously discussed phase I studies of trifluridine/tipiracil plus irinotecan in mCRCs are encouraging and suggest that trifluridine/tipiracil in combination with irinotecan may have better clinical activity in advanced BTCs than trifluridine/tipiracil alone.

## 1.4 Study Design

This is a single-arm, phase 2 trial to assess the efficacy of trifluridine/tipiracil plus irinotecan in advanced, refractory BTCs. The primary endpoint of this study is 16-week PFS rate. If 30% of patients remain progression-free at 16-weeks, this trial will be considered a success warranting bigger trials. A two-stage phase II design will be utilized. In the first stage, 15 patients will be enrolled. If 2 or more patients are progression-free and alive at 16 weeks, additional 10 patients will be enrolled. If 5 or fewer patients out of 25 evaluable patients remain progression-free at 16 weeks then the regimen will be considered ineffective. The total sample size of this study is 28 to account for 3 possible non-evaluable subjects. Patient will receive trifluridine/tipiracil at the dose of 25 mg/m<sup>2</sup> on Days 1-5 and irinotecan 180 mg/m<sup>2</sup> on Day 1 of each 14-day cycle. Patient will receive treatment until disease progression or unacceptable toxicities. Patients will undergo restaging scans every 4 cycles. Subjects will be monitored for adverse events from the beginning of the study drug to 28 days after the last dose. We will collect blood samples for determination of cell-free DNA (cfDNA) and circulating tumor cells (CTCs) at baseline, after 4 cycles and at progression. We will collect tumor biopsy specimens before treatment initiation to develop patient-derived tumor organoid.

MC1941 8 MCCC Amendment 1



#### 2.0 Goals

## 2.1 Primary Goal

Determine the efficacy of trifluridine/tipiracil in combination with irinotecan in patients with refractory biliary tract cancers using progression-free survival (PFS) at 16 weeks.

## 2.2 Secondary Goals

- 2.21 Assess the safety and tolerability of trifluridine/tipiracil in combination with irinotecan in patients with refractory biliary tract cancers through adverse event monitoring.
- 2.22 Further explore the efficacy of trifluridine/tipiracil in combination with irinotecan in patients with refractory biliary tract cancers by overall response rates (ORR), disease control rates (DCR), and overall survival (OS).

#### 2.3 Correlative Research

- 2.31 To determine if the number of circulating tumor cells (CTCs) or the level of cell-free DNA (cfDNA) at baseline is prognostic or predictive to the response to therapy.
- 2.32 To determine if changes in CTCs or cfDNA correlate with efficacy endpoints.
- 2.33 To determine if drug response from a parallel *ex vivo* trial using patient-derived tumor organoid correlates with clinical response to trifluridine/tipiracil plus irinotecan
- 2.34 To evaluate the role of thymidine kinase 1 (TK1) in predicting the clinical benefit of trifluridine/tipiracil plus irinotecan and discover potential mechanisms of resistance using patient-derived tumor organoid and pre-treatment biopsy specimen.

## 2.4 Exploratory Research

2.41 To evaluate patients who received prior treatment with 5-FU independently from the entire population in the following areas: PFS, safety and tolerability, ORR, DCR, and OS.

## 3.0 Registration Patient Eligibility

- 3.1 Registration Inclusion Criteria
  - 3.11 Age  $\geq$ 18 years
  - 3.12 Histological confirmation of advanced biliary tract cancers including cancers originating in the gallbladder who have received at least one line of systemic anticancer therapy.

Note: Patients who have either progressed on or are intolerant to the prior therapy can be included in this study.

3.13 Measurable disease as defined by RECIST criteria (See Section 11.0)

NOTE: Tumor lesions in a previously irradiated area are not considered measurable disease. Disease that is measurable by physical examination only is not eligible.

- 3.14 ECOG Performance Status (PS) of 0 or 1 (Appendix I).
- 3.15 The following laboratory values obtained ≤21 days prior to registration.
  - Absolute neutrophil count (ANC) ≥1500/mm<sup>3</sup>
  - Platelet count  $\geq 100,000/\text{mm}^3$
  - Total bilirubin  $\leq 1.5 \times$  upper limit of normal (ULN)
  - Aspartate transaminase (AST) or alanine transaminase (ALT)  $\leq 3 \times ULN$
  - Creatinine  $\leq 1.5 \times ULN$
- 3.16 Negative pregnancy test done ≤7 days prior to registration, for persons of childbearing potential only.
- 3.17 Provide written informed consent.
- 3.18 Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study).
- 3.19 Willingness to provide mandatory blood and tissue specimens for correlative research (see Sections 14.0 and 17.0).

## 3.2 Registration - Exclusion criteria

- 3.21 Any of the following because this study involves an agent that has potential genotoxic, mutagenic and teratogenic effects:
  - Pregnant persons
  - Nursing persons
  - Persons of childbearing potential who are unwilling to employ adequate contraception for at least 3 months after the last dose of the study drug
- 3.22 Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
- 3.23 Immunocompromised patients and patients known to be HIV positive and currently receiving antiretroviral therapy.NOTE: Patients known to be HIV positive, but without clinical evidence of an

immunocompromised state, are eligible for this trial.

- 3.24 Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
- 3.25 Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm ≤21 days prior to registration.
- 3.26 Receiving any anticancer therapy for biliary tract cancer ≤21 days prior to registration.
- 3.27 Other active malignancy requiring treatment in ≤6 months prior to registration. EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix. NOTE: If there is a history of prior malignancy, they must not be receiving other specific treatment for their cancer.
- 3.28 History of myocardial infarction ≤6 months prior to registration, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias.
- 3.29 Previous treatment with irinotecan or irinotecan-based chemotherapy for biliary tract cancers.

#### 4.0 Test Schedule

#### 4.1 Test schedule for BTCs

| | Active Monitoring Phase | | | | | |
|---|---|---|---|---|---|---|
| | ≤21 days | Prior to | D1 of | | | Safety follow-up: |
| | prior to | C1D1 | each | Every 4 | End of | 30 days post |
| Tests and procedures <sup>1</sup> | registration | Tx | cycle | cycles | treatment | treatment |
| Window | | | ±7 days | ±7 days | ±7 days | ±7 days |
| History and exam, Wt, PS | X | | X | | X | X |
| Height | X | | | | | |
| Adverse event assessment | X | | X | | X | X |
| Pregnancy test <sup>2</sup> | X | | | | | |
| Hematology group:<br>CBC with differential | X | | X | | X | X |
| Chemistry group <sup>3</sup> | X | | X | | X | X |
| CA19-9 | | $X^4$ | | $X^5$ | X | |
| Tumor measurement <sup>6</sup> | $X^7$ | | | $X^8$ | X | |
| Tumor biopsy | | $X^{9R}$ | | | | |
| Research blood specimens | | X | $X^{10}$ | | X | |
| (see Section 14.0) <sup>10R</sup> | | Λ | Λ | | Λ | |
| Research tissue specimens | | X | | | | |
| (see <u>Section 17.0</u> ) <sup>11R</sup> | | Λ | | | | |
| Patient medication diary | | | X | | X | |
| (Appendix II) <sup>12</sup> | | | Λ | | Λ | |

Cycle = 14 days

R Research funded (see Section 19.0)

<sup>1</sup> All tests and procedures should be performed as needed for clinical care at treating physician's discretion.

Protocol Version Date: 14Apr2020

<sup>&</sup>lt;sup>2</sup> For persons of childbearing potential only: Must be done ≤7 days prior to registration.

<sup>&</sup>lt;sup>3</sup> Chemistry: albumin, alkaline phosphatase, AST, ALT, total and direct bilirubin, creatinine, potassium, sodium

<sup>&</sup>lt;sup>4</sup> Baseline prior to Cycle 1, Day 1, then every 4 cycles or as clinically indicated

<sup>&</sup>lt;sup>5</sup> To be performed ≤7 days prior to planned Day 1 of Cycles 5, 9, etc., or as clinically indicated

<sup>&</sup>lt;sup>6</sup> To be performed per Mayo Clinic institutional guidelines – suggest CT (chest, abdomen, and pelvis) or CT (chest) and MRI (abdomen, pelvis)

<sup>&</sup>lt;sup>7</sup> Can be performed ≤28 days prior to registration

<sup>&</sup>lt;sup>8</sup> To be performed ≤7 days prior to planned Day 1 of Cycles 5, 9, etc., or as clinically indicated

<sup>&</sup>lt;sup>9</sup> Research biopsy after registration and prior to treatment on C1D1. Research biopsy may be omitted after discussion with PI, if it is not medically feasible or exceeds lab capacity.

<sup>&</sup>lt;sup>10</sup> Research blood specimens to be collected on Cycle 1 Day 1 (or any time between registration and Cycle 1 Day 1), Cycle 3 Day 1 and end of treatment (see Section 14.0)

<sup>&</sup>lt;sup>11</sup> Research tissue specimens to be collected during research biopsy any time between registration and prior to treatment on C1D1 (see Section 17.0). Biopsy can be omitted for patients for whom investigator deems it unsafe.

<sup>&</sup>lt;sup>12</sup> The diary must begin the day the patient starts taking the medication, and must be completed per protocol and returned to the treating institution at each visit.

## 4.2 Event Monitoring/Survival Follow-up

| | | Event Monitoring Phase <sup>1</sup> | | | |
|---|---|---|---|---|---|
| | q. 3 | | | | |
| | months | | After PD | | |
| | until PD | At PD | q. 3 months | Death | New Primary |
| Event monitoring | X | X | X | X | At each occurrence |

1. If a patient is still alive 2 years after registration, no further follow-up is required.

## 5.0 Stratification Factors OR Grouping Factor: None

## **6.0** Registration Procedures

## 6.1 Registration (Step 1):

To register a patient, access the Mayo Clinic Cancer Center (MCCC) web page and enter the registration/randomization application. The registration/ randomization application is available 24 hours a day, 7 days a week. Back up and/or system support contact information is available on the website. If unable to access the website, call the MCCC Registration Office at (507) 284-2753 between the hours of 8 a.m. and 4:30 p.m. Central Time (Monday through Friday).

The instructions for the registration/randomization application are available on the MCCC web page and detail the process for completing and confirming patient registration. Prior to initiation of protocol treatment, this process must be completed in its entirety and an MCCC subject ID number must be available as noted in the instructions. It is the responsibility of the individual registering the patient to confirm the process has been successfully completed prior to release of the study agent. Patient registration via the registration/randomization application can be confirmed in any of the following ways:

- Refer to "Instructions for Remote Registration" in section "Finding/Displaying Information about A Registered Subject."

## 6.2 Verification of materials

Prior to accepting the registration, registration/randomization application will verify the following:

- IRB approval at the registering institution
- Patient eligibility
- Existence of a signed consent form
- Existence of a signed authorization for use and disclosure of protected health information

## 6.3 Documentation of IRB approval

Documentation of IRB approval must be on file in the Registration Office before an investigator may register any patients.

In addition to submitting initial IRB approval documents, ongoing IRB approval documentation must be on file (no less than annually) at the Registration Office If the necessary documentation is not submitted in advance of attempting

patient registration, the registration will not be accepted and the patient may not be enrolled in the protocol until the situation is resolved.

When the study has been permanently closed to patient enrollment, submission of annual IRB approvals to the Registration Office is no longer necessary.

## 6.4 Correlative Research

## 6.41 Mandatory

A mandatory correlative research component is part of this study, the patient will be automatically registered onto this component (see Sections 3.19, 14.0 and 17.0).

## 6.42 Banking

At the time of registration, the following will be recorded:

- Patient has/has not given permission to store and use his/her sample(s) for future research on cancer at Mayo Clinic.
- Patient has/has not given permission to store and use his/her sample(s) for future research to learn, prevent, or treat other health problems.
- Patient has/has not given permission for MCCC to give his/her sample(s) to researchers at other institutions.

## 6.5 Treatment on protocol

Treatment on this protocol must commence at Mayo Clinic under the supervision of a medical oncologist.

#### 6.6 Treatment start

Treatment cannot begin prior to registration and must begin ≤14 days after registration.

#### 6.7 Pretreatment

Pretreatment tests/procedures (see <u>Section 4.0</u>) must be completed within the guidelines specified on the test schedule.

## 6.8 Baseline symptoms

All required baseline symptoms (see Section 10.6) must be documented and graded.

## 6.9 Study Conduct

The clinical trial will be conducted in compliance with regulations (21 CFR 312, 50, and 56), guidelines for Good Clinical Practice (ICH Guidance E6), and in accordance with general ethical principles outlined in the Declaration of Helsinki; informed consent will be obtained from all participating patients; the protocol and any amendments will be subject to approval by the designated IRB prior to implementation, in accordance with 21 CFR 56.103(a); and subject records will be stored in a secure location and subject confidentiality will be maintained. The investigator will be thoroughly familiar with the appropriate use of the study drug as described in the protocol and Investigator's Brochure. Essential clinical documents will be maintained to demonstrate the validity of the study and the integrity of the data collected. Master files should be established at the beginning of the study, maintained for the duration of the study and retained according to the appropriate regulations.

## 7.0 Protocol Treatment

#### 7.1 Treatment Schedule

All patients will receive study medication trifluridine/tipiracil (FTD/TPI) with irinotecan in a 14-day treatment cycle. Trifluridine/tipiracil is available in 15 and 20 mg tablets. Study medication should be administered as outlined in the protocol.

Use actual weight or estimated dry weight if fluid retention. BSA needs to be rounded to 2 decimal places. The study medication needs to be stored at the room temperature.

Trifluridine/tipiracil is administered in 14-day cycles. The starting dose of trifluridine/tipiracil is 25 mg/m². The study drug will be administered on Days 1-5 of 14-day cycle. If a patient starts treatment in the afternoon on Day 1 and can't take the morning dose of trifluridine/tipiracil, patient will take trifluridine/tipiracil on the morning on Day 6. This will allow patients to receive full dose of the therapy. No additional doses of trifluridine/tipiracil will be made up through the treatment cycle.

Irinotecan is administered in 14-day cycles. The starting dose of irinotecan is 180 mg/m<sup>2</sup>. It will be administered on Day 1 of 14-day cycle.

#### 7.11 Treatment medication table

| Agent | Route | Day | Starting Dose |
|---|---|---|---|
| Trifluridine/tipiracil (FTD/TPI) | PO | 1-5 | 25 mg/m <sup>2</sup> /dose twice daily |
| Irinotecan | IV | 1 | 180 mg/m <sup>2</sup> /dose once |
| None | | 6-14 | No treatment |

Cycle = 14 days

NOTE: On days when irinotecan and FTD/TPI are both administered, prefer morning dose of FTD/TPI taken in the clinic, if possible

## 7.12 Trifluridine/tipiracil dose calculation based on BSA

| Trifluridine/tipiracil dose | | Dosage in mg | Tablets per dose | |
|---|---|---|---|---|
| (twice daily) | BSA (m <sup>2</sup> ) | (twice daily) | 15 mg | 20 mg |
| $25 \text{ mg/m}^2$ | <1.10 | 25 <sup>a</sup> | 2 (PM) <sup>a</sup> | $1 (AM)^a$ |
| $25 \text{ mg/m}^2$ | 1.10-1.29 | 30 | 2 | 0 |
| $25 \text{ mg/m}^2$ | 1.30-1.49 | 35 | 1 | 1 |
| $25 \text{ mg/m}^2$ | 1.50-1.69 | 40 | 0 | 2 |
| $25 \text{ mg/m}^2$ | 1.70-1.89 | 45 | 3 | 0 |
| $25 \text{ mg/m}^2$ | 1.90-2.09 | 50 | 2 | 1 |
| $25 \text{ mg/m}^2$ | 2.10-2.29 | 55 | 1 | 2 |
| $25 \text{ mg/m}^2$ | ≥2.30 | 60 | 0 | 3 |

<sup>&</sup>lt;sup>a</sup> At a total daily dose of 50 mg, patients should take  $1 \times 20$ -mg tablet in the morning and  $2 \times 15$ -mg tablets in the evening.

#### 7.13 Irinotecan

Irinotecan dose calculation is based on BSA per institutional standards. Irinotecan should be given IV per institutional standards. Package insert recommended infusion time is 90 minutes.

NOTE: On days when irinotecan and FTD/TPI are both administered, prefer morning dose of FTD/TPI is taken in the clinic, if possible.

## 7.2 Self-administration statement for FTD/TPI

Patients can be instructed in administration techniques and granted treatment independence. Any missed doses will be recorded. Patients will be instructed to:

- Store the study medication at room temperature
- Take the study medication on schedule
- Report any missed doses
- Take study medication within 1 hour after completing morning or evening meals with a glass of water
- If the patient vomits after taking the study medication, the dose should not be replaced.
- Return the unused medication at end of every cycle.
- If a patient forgets to take a dose (morning or evening), the missed dose should not be made up

## 7.3 Treatment by local medical doctor (LMD)

Treatment by a local medical doctor (LMD) is <u>not</u> allowed on this study.

## 7.4 Discontinuation of study treatment

Study treatment will be discontinued for any of the following:

- Disease progression
- Unacceptable adverse events
- Non-compliance (need to be discussed with PI)
- Withdrawal of consent by the patient
- Provider's discretion for patient's best interest (need to be discussed with PI)

In rare circumstances, patient can be continued beyond progression if the investigator determines that patient is benefitting from the treatment. This decision will need to be made in conjunction with PI and will be only allowed in exceptional circumstances.

## 8.0 Dosage Modification Based on Adverse Events

For the first two cycles, strictly follow the modifications in this table. Thereafter, these modifications should be regarded as guidelines to produce mild-to-moderate, but not debilitating, side effects. Under exceptional circumstances, at the investigator discretion (in consultation with principal investigator) dose modifications or treatment interruption or continuation can be considered if it's considered to be in the best interest of a patient. If multiple adverse events are seen, administer dose based on greatest reduction required for any single adverse event observed. Reductions apply to treatment given in the preceding cycle and are based on adverse events observed since the prior dose. The criteria for dose modifications of trifluridine/tipiracil or irinotecan for toxicities will be considered if an adverse event is at least possibly related to trifluridine/tipiracil or irinotecan. Dose modification will be done only for study drug related adverse event only.

If either drug is delayed for more than 28 days due to adverse event possibly, probably, or definitely related to study drug, then discontinue that drug

If one drug is discontinued due to adverse events, the patient continues on trial on the other drug. If both drugs are discontinued, the patient goes to event monitoring.

NCI Common Terminology Criteria for Adverse Events (CTCAE) current version 5.0\* will be utilized for dose modification unless otherwise specified. Up to three dose level reductions are allowed. Once reduced for an adverse event, no increase in dose of trifluridine/tipiracil will be allowed.

\* Located at

#### Definitions:

- > Omit = The current dose(s) for the specified drug(s) during a cycle is skipped. The patient does not make up the omitted dose(s) at a later time.
- ➤ Hold/Delay = The current dose(s) of all drugs during a cycle is delayed. The patient does make up the delayed dose(s) when the patient meets the protocol criteria to restart drugs.
- ➤ **Discontinue** = The specified drug(s) are totally stopped.
- 8.1 Dose Levels (Based on Adverse Events in Tables 8.2 and 8.3)

| Dose Level | Trifluridine/tipiracil (FTD/TPI) | Irinotecan |
|------------|----------------------------------|-----------------------------|
| 0* | 25 mg/m <sup>2</sup> /dose BID | 180 mg/m <sup>2</sup> /dose |
| -1 | 25 mg/m <sup>2</sup> /dose BID | 150 mg/m <sup>2</sup> /dose |
| -2 | 20 mg/m <sup>2</sup> /dose BID | 150 mg/m <sup>2</sup> /dose |
| -3 | 20 mg/m <sup>2</sup> /dose BID | 120 mg/m <sup>2</sup> /dose |

<sup>\*</sup>Dose level 0 refers to the starting dose.

**NOTE:** Adverse events requiring a dose-reduction step for any or all drugs beyond the three dose-reduction steps (levels -1, -2 and -3) will be at the discretion of the treating physician, if the decision is made for the patient to be kept on study. These dose reductions must be clearly recorded in reported clinical data.

NOTE: Permanently discontinue FTD/TPI in patients unable to tolerate a dose of 20 mg/m<sup>2</sup> PO BID.

| 8.11 | Trifluridine/tipiraci | l dose calculation aft | er dose modifications | based on BSA |
|---|---|---|---|---|

| Trifluridine/tipiracil dose | | Dosage in mg | Tablets | per dose |
|---|---|---|---|---|
| (twice daily) | BSA (m <sup>2</sup> ) | (twice daily) | 15 mg | 20 mg |
| $20 \text{ mg/m}^2$ | <1.14 | 20 | 0 | 1 |
| $20 \text{ mg/m}^2$ | 1.14-1.34 | 25ª | 2 (PM) <sup>a</sup> | 1 (AM) <sup>a</sup> |
| $20 \text{ mg/m}^2$ | 1.35-1.59 | 30 | 2 | 0 |
| $20 \text{ mg/m}^2$ | 1.60-1.94 | 35 | 1 | 1 |
| $20 \text{ mg/m}^2$ | 1.95-2.09 | 40 | 0 | 2 |
| $20 \text{ mg/m}^2$ | 2.10-2.29 | 45 | 3 | 0 |
| $20 \text{ mg/m}^2$ | ≥2.30 | 50 | 2 | 1 |

<sup>&</sup>lt;sup>a</sup> For the total daily dose of 50 mg, patients should take  $1 \times 20$ -mg tablet in the morning and  $2 \times 15$ -mg tablets in the evening.

- 8.2 Dose Modifications Based on **Interval** Adverse Events (occurring within a cycle of treatment)
  - 8.21 For non-specified adverse events following criteria for dose modification will be used for adverse events occurring during the cycle:

| CTCAE | |
|-----------------------------|-------------------------------------------|
| Adverse Events <sup>1</sup> | ACTION |
| Grade 1 or 2 | Treat as scheduled |
| | Omit treatment until resolved to ≤Grade 2 |
| Grade 3 or 4 | If any Reduce the dose of FTD/TPI by one |
| | dose level |

<sup>&</sup>lt;sup>1</sup> Except for anemia, alopecia, clinically insignificant laboratory abnormalities, and inadequately treated nausea, vomiting, and diarrhea.

8.22 For specified adverse events the following criteria for dose modification will be used for adverse events occurring during the cycle:

| CTCAE | CTCAE | |
|---|---|---|
| System/Organ Class | Adverse Events | ACTION |
| Investigations | >( ÷rade / | Omit treatment for the duration of the cycle |
| Investigations | Platelet count decreased<br>≥Grade 3<br><50,000/mm <sup>3</sup> | Omit treatment for the duration of the cycle |

G-CSF can be used in this trial at the discretion of treating physician (see Section 9.2)

- 8.3 Dose Modifications at the **Time of Retreatment** (Beginning of a new cycle)
  - 8.31 The dose modification guidelines for non-specified adverse events on Day 1 of each cycle of the treatment are mentioned below:

| CTCAE Adverse Events <sup>1</sup> | ACTION |
|---|---|
| Grade 1 or 2 | Treat as scheduled |
| | Delay treatment until resolved to ≤Grade 2<br>Reduce the dose of both drugs by one dose level |

<sup>&</sup>lt;sup>1</sup> Except for anemia, alopecia, clinically insignificant laboratory abnormalities, and inadequately treated nausea, vomiting, and diarrhea.

8.32 The dose modification guidelines for specified adverse events on Day 1 of each cycle of the treatment are mentioned below:

| CTCAE | CTCAE | |
|---|---|---|
| System/Organ Class | <b>Adverse Events</b> | ACTION |
| Blood and lymphatic system disorders | Febrile<br>neutropenia<br>(≥Grade 3) | Delay treatment by 1 week (see Section 9.0 for supportive care guidelines) If resolved within 1 week (7 days), retreat at same dose Reduce dose by one dose level of both drugs for next treatment only if there is more than one week delay in start of next cycle |
| Investigations | Neutrophil count<br>decreased<br>≥Grade 2<br><1500/mm <sup>3</sup> | Delay treatment by 1 week (see Section 9.0 for supportive care guidelines) If resolved to ≤Grade 1 within 1 week (7 days), retreat at same dose Reduce dose by one dose level of both drugs for next treatment only if there is more than one week delay in start of next cycle |
| Investigations | Platelet count<br>decreased<br><75,000/mm <sup>3</sup> | Delay treatment by 1 week(see Section 9.0 for supportive care guidelines) If resolved to ≤Grade 1 within 1 week (7 days), retreat at same dose Reduce dose by one dose level of both drugs for next treatment only if there is more than one week delay in start of next cycle |

## 9.0 Ancillary Treatment/Supportive Care

## 9.1 Full supportive care

Patients should receive full supportive care while on this study. This includes blood product support, antibiotic treatment, and treatment of other newly diagnosed or concurrent medical conditions. All blood products and concomitant medications such as antidiarrheals, analgesics, and/or antiemetics received from the first day of study treatment administration until 30 days after the final dose will be recorded in the medical records.

## 9.2 Blood products and growth factors

Blood products and growth factors should be utilized as clinically warranted and following institutional policies and recommendations. The use of growth factors should follow published guidelines of the Journal of Clinical Oncology, Volume 33, No 28 (October 1), 2015: pp. 3199-3212 (WBC growth factors) AND Journal of Clinical Oncology, Volume 28, No 33 (November 20), 2010: pp. 4955-5010 (darbepoetin/epoetin).

## 9.3 Antiemetics

Antiemetics may be used at the discretion of the attending physician.

#### 9.4 Diarrhea

Diarrhea could be managed conservatively with loperamide. The recommended dose of loperamide is 4 mg at first onset, followed by 2 mg every 2-4 hours until diarrhea free (maximum 16 mg/day).

In the event of Grade 3 or 4 diarrhea, the following supportive measures are allowed: hydration, octreotide, and antidiarrheals.

If diarrhea is severe (requiring intravenous rehydration) and/or associated with fever or severe neutropenia (Grade 3 or 4), broad-spectrum antibiotics must be prescribed. Patients with severe diarrhea or any diarrhea associated with severe nausea or vomiting **should be hospitalized** for intravenous hydration and correction of electrolyte imbalances.

## 10.0 Adverse Event (AE) Monitoring and Reporting

The site principal investigator is responsible for reporting any/all serious adverse events to the sponsor as described within the protocol, regardless of attribution to study agent or treatment procedure.

The sponsor/sponsor-investigator is responsible for notifying FDA and all participating investigators in a written safety report of any of the following:

- Any suspected adverse reaction that is both serious and unexpected.
- Any findings from laboratory animal or *in vitro* testing that suggest a significant risk for human subjects, including reports of mutagenicity, teratogenicity, or carcinogenicity.
- Any findings from epidemiological studies, pooled analysis of multiple studies, or clinical studies, whether or not conducted under an IND and whether or not conducted by the sponsor, that suggest a significant risk in humans exposed to the drug
- Any clinically important increase in the rate of a serious suspected adverse reaction over the rate stated in the protocol or Investigator's Brochure (IB).

Summary of SAE Reporting for this study (please read entire section for specific instructions):



## **Definitions**

Adverse Event

Any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related.

MC1941 21 MCCC Amendment 1

## Suspected Adverse Reaction

Any adverse event for which there is a reasonable possibility that the drug caused the adverse event.

## **Expedited Reporting**

Events reported to sponsor within 24 hours, 5 days or 10 days of study team becoming aware of the event.

#### Routine Reporting

Events reported to sponsor via case report forms

## Events of Interest

Events that would not typically be considered to meet the criteria for expedited reporting, but that for a specific protocol are being reported via expedited means in order to facilitate the review of safety data (may be requested by the FDA or the sponsor).

## Unanticipated Adverse Device Event (UADE)

Any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, a device, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan or application (including a supplementary plan or application), or any other unanticipated serious problem associated with a device that relates to the rights, safety, or welfare of subjects.

#### 10.1 Adverse Event Characteristics

CTCAE term (AE description) and grade: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for AE reporting. All appropriate treatment areas should have access to a copy of the CTCAE version 5.0. A copy of the CTCAE version 5.0 can be downloaded from the CTEP web site:

- a. Identify the grade and severity of the event using the CTCAE version 5.0.
- b. Determine whether the event is expected or unexpected (see Section 10.2).
- c. Determine if the adverse event is related to the study intervention (agent, treatment or procedure) (see Section 10.3).
- d. Determine whether the event must be reported as an expedited report. If yes, determine the timeframe/mechanism (see Section 10.4).
- e. Determine if other reporting is required (see Section 10.5).
- f. Note: All AEs reported via expedited mechanisms must also be reported via the routine data reporting mechanisms defined by the protocol (see Sections 10.6 and 18.0).

NOTE: A severe AE is NOT the same as a serious AE, which is defined in Section 10.4.

## 10.2 Expected vs. Unexpected Events

Expected events - are those described within the Section 15.0 of the protocol, the study specific consent form, package insert (if applicable), and/or the investigator brochure, (if an investigator brochure is not required, otherwise described in the general investigational plan).

*Unexpected adverse events* or suspected adverse reactions are those not listed in Section 15.0 of the protocol, the study specific consent form, package insert (if applicable), or in the investigator brochure (or are not listed at the specificity or severity that has been observed); if an investigator brochure is not required or available, is not consistent with

the risk information described in the general investigational plan.

*Unexpected* also refers to adverse events or suspected adverse reactions that are mentioned in the investigator brochure as occurring with a class of drugs but have not been observed with the drug under investigation.

An investigational agent/intervention might exacerbate the expected AEs associated with a commercial agent. Therefore, if an expected AE (for the commercial agent) occurs with a higher degree of severity or specificity, expedited reporting is required.

NOTE: \*The consent form may contain study specific information at the discretion of the Principal Investigator; it is possible that this information may NOT be included in the protocol or the investigator brochure. Refer to protocol or IB for reporting needs.

## 10.3 Attribution to agent(s) or procedure

When assessing whether an adverse event (AE) is related to a medical agent(s) medical or procedure, the following attribution categories are utilized:

Definite - The AE is clearly related to the agent(s)/procedure.

Probable - The AE *is likely related* to the agent(s)/procedure.

Possible - The AE may be related to the agent(s)/procedure.

Unlikely - The AE is doubtfully related to the agent(s)/procedure.

Unrelated - The AE is clearly NOT related to the agent(s)/procedure.

## 10.31 AEs Experienced Utilizing Investigational Agents and Commercial Agent(s)

**NOTE:** When a commercial agent(s) is (are) used on the same treatment arm as the investigational agent/intervention (also, investigational drug, biologic, cellular product, or other investigational therapy under an IND), the **entire combination (arm) is then considered an investigational intervention for reporting**.

- An AE that occurs on a combination study must be assessed in accordance with the guidelines for investigational agents/interventions.
- An AE that occurs prior to administration of the investigational agent/intervention
  must be assessed as specified in the protocol. In general, only Grade 4 and 5 AEs
  that are unexpected with at least possible attribution to the commercial agent require
  an expedited report, unless hospitalization is required. Refer to Section 10.4 for
  specific AE reporting requirements or exceptions.

An investigational agent/intervention might exacerbate the expected AEs associated with a commercial agent. Therefore, if an expected AE (for the commercial agent) occurs with a higher degree of severity or specificity, expedited reporting is required.

- An increased incidence of an expected adverse event (AE) is based on the
  patients treated for this study at their site. A list of known/expected AEs is
  reported in the package insert or the literature, including AEs resulting from a
  drug overdose.
- Commercial agent expedited reports must be submitted to the FDA via MedWatch 3500A for Health Professionals (complete all three pages of the form).



Instructions for completing the MedWatch 3500A:

10.32 EXPECTED Serious Adverse Events: Protocol Specific Exceptions to Expedited Reporting

For this protocol only, the following Adverse Events/Grades are expected to occur within this population and do not require Expedited Reporting. These events must still be reported via Routine Reporting (see Section 10.6).\*

\*Report any clinically important increase in the rate of a serious suspected adverse reaction (at your study site) over that which is listed in the protocol or investigator brochure as an expedited event.

\*Report an expected event that is greater in severity or specificity than expected as an expedited event.

| CTCAE | | CTCAE Grade at which the |
|---|---|---|
| System Organ Class | | event will not be reported in |
| (SOC) | Adverse event/ Symptoms | an expedited manner <sup>1</sup> |
| Blood and lymphatic system disorders | | |
| Gastrointestinal disorders | Diarrhea | ≤Grade 3 |
| | Nausea | ≤Grade 3 |
| | Vomiting | ≤Grade 3 |
| General disorders and | Fatigue | ≤Grade 3 |
| administrations site conditions | Malaise | ≤Grade 3 |
| Investigations | Lymphocyte count decreased | ≤Grade 4 |
| | Neutrophil count decreased | ≤Grade 4 |
| | Platelet count decreased | ≤Grade 4 |
| | White blood cell count decreased | ≤Grade 4 |

<sup>&</sup>lt;sup>1</sup> These exceptions only apply if the adverse event does not result in hospitalization. If the adverse event results in hospitalization, then the standard expedited adverse events reporting requirements must be followed.

Specific protocol exceptions to expedited reporting should be reported expeditiously by investigators **ONLY** if they exceed the expected grade of the event.

The following hospitalizations are not considered to be SAEs because there is no "adverse event" (*i.e.*, there is no untoward medical occurrence) associated with the hospitalization:

- Hospitalizations for respite care
- Planned hospitalizations required by the protocol
- Hospitalization planned before informed consent (where the condition requiring the hospitalization has not changed post study drug administration)
- Hospitalization for elective procedures unrelated to the current disease and/or treatment on this trial
- Hospitalization for administration of study drug or insertion of access for administration of study drug
- Hospitalization for routine maintenance of a device (e.g., battery replacement) that was in place before study entry
- Hospitalization, or other serious outcomes for signs and symptoms of progression of the cancer.

## 10.4 Expedited Reporting Requirements for IND Agents

10.41 Phase 1 and Early Phase 2 Studies: Expedited Reporting Requirements for Adverse Events that Occur on Studies under an IND within 30 Days of the Last Administration of the Investigational Agent/Intervention 1,2

## FDA REPORTING REQUIREMENTS FOR SERIOUS ADVERSE EVENTS (21 CFR Part 312)

NOTE: Investigators <u>MUST</u> immediately report to the sponsor <u>ANY</u> Serious Adverse Events, whether or not they are considered related to the investigational agent(s)/intervention (21 CFR 312.64)

An adverse event is considered serious if it results in ANY of the following outcomes:

- 1) Death
- 2) A life-threatening adverse event
- An adverse event that results in inpatient hospitalization or prolongation of existing hospitalization for ≥ 24 hours
- 4) A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- 5) A congenital anomaly/birth defect.
- 6) Important Medical Events (IME) that may not result in death, be life threatening, or require hospitalization may be considered serious when, based upon medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. (FDA, 21 CFR 312.32; ICH E2A and ICH E6).

<u>ALL SERIOUS</u> adverse events that meet the above criteria MUST be immediately reported to the sponsor within the timeframes detailed in the table below.

| Hospitalization | Grade 1 and Grade 2 Timeframes | Grade 3-5<br>Timeframes |
|---|---|---|
| Resulting in<br>Hospitalization<br>≥24 hrs | 7 Calendar Days | 24-Hour 3 Calendar |
| Not resulting in<br>Hospitalization<br>≥24 hrs | Not required | Days |

#### **Expedited AE reporting timelines are defined as:**

- "24-Hour; 3 Calendar Days" The AE must initially be reported within 24 hours of learning of the AE, followed by a complete expedited report within 3 calendar days of the initial 24-hour report.
- "7 Calendar Days" A complete expedited report on the AE must be submitted within 7 calendar days of learning of the AE.

All Grade 3, 4, and Grade 5 AEs

## Expedited 7 calendar day reports for:

Grade 2 AEs resulting in hospitalization or prolongation of hospitalization

Effective Date: May 5, 2011

NOTE: Refer to Section 10.32 for exceptions to Expedited Reporting

<sup>&</sup>lt;sup>1</sup>Serious adverse events that occur more than 30 days after the last administration of investigational agent/intervention and have an attribution of possible, probable, or definite require reporting as follows: Expedited 24-hour notification followed by complete report within 3 calendar days for:

<sup>&</sup>lt;sup>2</sup> For studies using PET or SPECT IND agents, the AE reporting period is limited to 10 radioactive half-lives, rounded UP to the nearest whole day, after the agent/intervention was last administered. Footnote "1" above applies after this reporting period.

## 10.42 General reporting instructions

The Mayo IND and/or MCCC Compliance will assist the sponsor-investigator in the processing of expedited adverse events and forwarding of suspected unexpected serious adverse reactions (SUSARs) to the FDA and IRB.

Use Mayo Expedited Event Report form

or investigational agents or commercial/investigational agents on the same arm and attach MedWatch 3500A.

Submit to NCCN via email

AND

Submit to Taiho Oncology Inc. Pharmacovigilance contact information for IIT sites to report SAEs (email preferred):

- FAX:
- Hotline phone: (phone number is only to ask questions, not to report SAEs)

## For commercial agents:

Submit form MedWatch 3500A to the FDA,

## Data Safety Update Requests (DSUR)

If requested by Institution, TAIHO shall provide the Institution with the final version of this DSUR report within 15 calendar days after submission to health agencies and ethics committees.

## 10.43 Reporting of re-occurring SAEs

ALL SERIOUS adverse events that meet the criteria outlined in table 10.41 MUST be immediately reported to the sponsor within the timeframes detailed in the corresponding table. This reporting includes, but is not limited to SAEs that re-occur again after resolution.

#### 10.5 Other Required Reporting

10.51 Unanticipated Problems Involving Risks to Subjects or Others (UPIRTSOS)

Unanticipated Problems Involving Risks to Subjects or Others (UPIRTSOS) in general, include any incident, experience, or outcome that meets **all** of the following criteria:

- 1. Unexpected (in terms of nature, severity, or frequency) given (a) the research procedures that are described in the protocol-related documents, such as the IRB-approved research protocol and informed consent document; and (b) the characteristics of the subject population being studied;
- 2. Related or possibly related to participation in the research (in this guidance document, possibly related means there is a reasonable possibility that the

incident, experience, or outcome may have been caused by the procedures involved in the research); and

Suggests that the research places subjects or others at a greater risk of harm (including physical, psychological, economic, or social harm) than was previously known or recognized.

Some unanticipated problems involve social or economic harm instead of the physical or psychological harm associated with adverse events. In other cases, unanticipated problems place subjects or others at increased *risk* of harm, but no harm occurs.

Note: If there is no language in the protocol indicating that pregnancy is not considered an adverse experience for this trial, and if the consent form does not indicate that subjects should not get pregnant/impregnate others, then any pregnancy in a subject/patient or a male patient's partner (spontaneously reported) which occurs during the study or within 120 days of completing the study should be reported as a UPIRTSO.

## Mayo Clinic Cancer Center (MCCC) Institutions:

If the event meets the criteria for IRB submission as a Reportable Event/UPIRTSO, provide the appropriate documentation and use the Mayo Clinic Cancer Center Expedited Event Report form

he Mayo Clinic Compliance Unit will review and process the submission to the Mayo Clinic IRB and work with the IND Coordinator for submission to FDA.

#### 10.52 Death

Note: A death on study requires both routine and expedited reporting regardless of causality, unless as noted below. Attribution to treatment or other cause must be provided.

Any death occurring within 30 days of the last dose, regardless of attribution to an agent/intervention under an IND requires expedited reporting within 24-hours.

Any death occurring greater than 30 days with an attribution of possible, probable, or definite to an agent/intervention under an IND requires expedited reporting within 24-hours.

## Reportable categories of Death

- Death attributable to a CTCAE term.
- Death Neonatal: A disorder characterized by cessation of life during the first 28 days of life.
- Death NOS: A cessation of life that cannot be attributed to a CTCAE term associated with Grade 5.
- Sudden death NOS: A sudden (defined as instant or within one hour of the onset of symptoms) or an unobserved cessation of life that cannot be attributed to a CTCAE term associated with Grade 5.
- Death due to progressive disease that cannot be attributed to a CTCAE term associated with Grade 5 should be reported as Grade 5 Disease

**progression** under the system organ class (SOC) of Gneral disorders and administration site conditions. Evidence that the death was a manifestation of underlying disease (e.g., radiological changes suggesting tumor growth or progression: clinical deterioration associated with a disease process) should be submitted.

## 10.53 Secondary Malignancy

- A *secondary malignancy* is a cancer caused by treatment for a previous malignancy (e.g., treatment with investigational agent/intervention, radiation or chemotherapy). A secondary malignancy is not considered a metastasis of the initial neoplasm.
- All secondary malignancies that occur following treatment with an agent under an IND will be reported. Three options are available to describe the event:
  - Neoplasms benign, malignant and unspecified, (incl cysts and polyps)
     Leukemia secondary to oncology chemotherapy (e.g., Acute Myeloctyic Leukemia [AML])
  - Neoplasms benign, malignant and unspecified, (incl cysts and polyps)
     Myelodysplastic syndrome (MDS)
  - Neoplasms benign, malignant and unspecified, (incl cysts and polyps)
     Treatment-related secondary malignancy
- Any malignancy possibly related to cancer treatment (including AML/MDS) should also be reported via the routine reporting mechanisms outlined in each protocol.

## 10.54 Second Malignancy

A second malignancy is one unrelated to the treatment of a prior malignancy (and is NOT a metastasis from the initial malignancy). Second malignancies require ONLY routine reporting unless otherwise specified.

## 10.55 Pregnancy, Fetal Death, and Death Neonatal

the child/fetus is the patient.

If a female subject (or female partner of a male subject) taking investigational product becomes pregnant, the subject taking should notify the Investigator, and the pregnant female should be advised to call her healthcare provider immediately. The patient should have appropriate follow-up as deemed necessary by her physician. If the baby is born with a birth defect or anomaly, a second expedited report is required.

Prior to obtaining private information about a pregnant woman and her infant, the investigator must obtain consent from the pregnant woman and the newborn infant's parent or legal guardian before any data collection can occur. A consent form will need to be submitted to the IRB for these subjects if a pregnancy occurs. If informed consent is not obtained, no information may be collected. In cases of fetal death, miscarriage or abortion, the mother is the patient. In cases where the child/fetus experiences a serious adverse event other than fetal death,

NOTE: When submitting Mayo Expedited Adverse Event Report reports for "Pregnancy", "Pregnancy loss", or "Neonatal loss", the potential risk of exposure of the fetus to the investigational agent(s) or chemotherapy agent(s) should be

documented in the "Description of Event" section. Include any available medical documentation. Include this form:

#### 10.551 Pregnancy

Pregnancy should be reported in an expedited manner as **Grade 3** "**Pregnancy**, **puerperium and perinatal conditions** - **Other** (**pregnancy**)" under the Pregnancy, puerperium and perinatal conditions SOC. Pregnancy should be followed until the outcome is known.

## 10.552 Fetal Death

Fetal death is defined in CTCAE as "A disorder characterized by death in utero; failure of the product of conception to show evidence of respiration, heartbeat, or definite movement of a voluntary muscle after expulsion from the uterus, without possibility of resuscitation."

Fetal loss at any gestational age should be reported expeditiously, as **Grade 4 "Pregnancy loss"** under the Pregnancy, puerperium and perinatal conditions SOC.

## 10.553 Death Neonatal

Neonatal death, defined in CTCAE as "Newborn death occurring during the first 28 days after birth" that is felt by the investigator to be at least possibly due to the investigational agent/intervention.

A neonatal death should be reported expeditiously as **Grade 4 "Death neonatal"** under the SOC of General disorders and administration site conditions

## 10.6 Required Routine Reporting

#### 10.61 Baseline and Adverse Events Evaluations

Pretreatment symptoms/conditions to be graded at baseline and adverse events to be graded at each evaluation.

Grading is per CTCAE v5.0 **unless** alternate grading is indicated in the table below:

| CTCAE<br>System/Organ/Class<br>(SOC) | Adverse event/Symptoms | Baseline | Each<br>evaluation |
|---|---|---|---|
| Blood and<br>lymphatic disorders | Anemia | X | X |
| Investigations | Neutrophil count decreased | X | X |
| | Platelet count decreased | X | X |

#### 10.62 All other AEs

Submit via appropriate MCCC Case Report Forms (i.e., paper or electronic, as applicable) the following AEs experienced by a patient and not specified in Section 10.6:

- 10.621 Grade 2 AEs deemed *possibly, probably, or definitely* related to the study treatment or procedure.
- 10.622 Grade 3 and 4 AEs regardless of attribution to the study treatment or procedure.
- 10.623 Grade 5 AEs (Deaths)
  - 10.6231 Any death within 30 days of the patient's last study treatment or procedure regardless of attribution to the study treatment or procedure.
  - 10.6232 Any death more than 30 days after the patient's last study treatment or procedure that is felt to be at least possibly treatment related must also be submitted as a Grade 5 AE, with a CTCAE type and attribution assigned.
- 10.7 Late Occurring Adverse Events

Refer to the instructions in the Forms Packet (or electronic data entry screens, as applicable) regarding the submission of late occurring AEs following completion of the Active Monitoring Phase (i.e., compliance with Test Schedule in Section 4.0).

10.8 Taiho Oncology Additional Event Reporting Instructions

For Investigators with an IND exemption:

## Reporting Clinical Safety Information to TAIHO

- a) The Physician shall monitor the Patient for adverse events and fulfil all the reporting requirements to FDA in accordance with Applicable Laws. The Physician shall also inform Taiho Oncology of serious adverse events:
  - § Unexpected Fatal or Life Threatening Suspected Adverse Reactions- Report to Taiho Oncology, Inc. within 24 hours
  - § Serious & Unexpected Suspected Adverse Reactions- Report to Taiho Oncology, Inc. within 24 hours.
  - § All other Serious cases (Expected and Related; Expected and Not related; Unexpected and Not related)- Report to Taiho Oncology within 2 weeks of awareness.
- b) All serious adverse events via a MedWatch Form need to be sent to the Taiho Oncology, Inc., via
- MedWatch reports must clearly specify SAE term(s) and corresponding investigator causality assessment.
- d) Taiho will send SUSARs to Regulatory Authorities via a MedWatch form within 7 Calendar Days for all fatal/life threatening events and 15 Calendar Days for all other serious events.

## Drug Exposure during Pregnancy and Lactation, or Paternal Drug Exposure Reports

The Institution will report Exposure During Pregnancy and Lactation, or Paternal Drug Exposure on any Clinical Trial Subject while participating in the Clinical Trial, and following exposure to a TAIHO IMP, to TAIHO (as specified below) using copies of the

original Pregnancy Report Form and within two weeks of first becoming aware of the pregnancy or exposure. If the partner of a Clinical Trial Subject becomes pregnant, the Institution may collect information about the pregnancy and birth if the partner agrees.

The Clinical Trial Subject will also be followed by the Institution to determine the outcome of the pregnancy (including any premature termination of the pregnancy). Information on the status of the mother and child will be forwarded to TAIHO. The Institution must provide final outcome of pregnancy to TAIHO. If any SAE(s) is observed in Clinical Trail Subject or fetus/child, then SAE(s) must also be reported to TAIHO following SAE Reporting guidelines.

# Routing of Drug Exposure during Pregnancy and Lactation, or Paternal Drug Exposure Reports

Such reports and Information as outlined above, including Investigator causality assessments against all concerned TAIHO IMP(s) and English translations where reporting Is from a non-English speaking country, shall be sent:

- by facsimile to PV CONTACT NUMBER:
- by e-mail to:

## Requesting Follow up information:

The institution will provide TAIHO with details of whom TAIHO shall address requests for follow up Information on SAE and pregnancy cases reported from this Clinical Trial, and further agree to update such contact details as necessary. At the time of this Agreement, all such requests should be addressed to: (ENTER INVESTIGATOR)

## SAE Reconciliation

Reconciliation shall be performed quarterly as an exchange of Line Listings or other means in English. On a quarterly basis, the institution shall provide to TAIHO a line listing or other means of cumulative SAE received to date. At the end of the Clinical Trial a global reconciliation shall be performed. Please reference contact information when sending this reconciliation. All serious adverse events via a MedWatch Form need to be sent to the FDA and to Taiho Oncology, Inc., via fax:

#### Additional Reporting Instructions for Taiho

Serious adverse events must be reported to Taiho Pharmacovigilance or designee within 24 hours from the time the investigator first becomes aware of the SAE. Comprehensive information available at the time of initial reporting (including narrative description, medical history and concomitant medications) needs to be provided with careful consideration regarding causality and serious criteria.

After the initial SAE notification to Taiho Pharmacovigilance or designee, follow-up SAE information will be submitted each time that important follow-up information (e.g., diagnosis, outcome, causality assessment, results of specific investigations) becomes available.

All SAEs **within** the follow-up window (e.g., within 30 days after the last dose of study drug or until the start of new antitumor therapy, whichever is earlier) established in the protocol will be reported to Taiho Pharmacovigilance or designee.

If serious medical occurrences including deaths **outside** the follow-up window established by the protocol are reported to or observed by the investigator that he/she believes are related to the administration of the investigational product, it is the investigator's responsibility to report this occurrence to Taiho Pharmacovigilance or designee.

## 10.81 Reporting of Deaths

All deaths occurring through the 30-day follow-up period must be reported to Taiho Pharmacovigilance or designee within 24 hours.

## 1. Death due to disease progression:

Disease progression (radiologic or clinical) with the outcome of death will not be reported as an SAE. However, relevant signs, symptoms and complications of disease progression (radiologic or clinical) must be reported as an AE or SAE if it meets the serious criteria. It should be indicated that the signs, symptoms and complications are related to disease progression.

#### 2. Death due to other causes:

Deaths due to reasons other than disease progression must be reported as an SAE.

Death is not an acceptable AE/SAE term. Death is an outcome of an SAE.

When reporting a death, the investigator will be required to identify which of the following best describes the category of death:

- Toxicity for study drugs
- Radiologic disease progression
- Clinical disease progression
- Other causes

## 10.82 Disease Progression

How to report events related to non-fatal disease progression:

- a. Disease progression is not an acceptable AE term. In cases of non-fatal disease progression, the relevant signs, symptoms and complications should be reported as an AE unless they meet the serious criteria. If any of the signs, symptoms and complications meets any of the serious criteria, they should be reported as an SAE. In both cases it should be indicated whether the signs, symptoms and complications are related to disease progression.
- b. Radiologic disease progression without relevant signs, symptoms and complications will **not** be reported as an AE or SAE.

#### 10.83 Pregnancy

If a patient becomes pregnant while in the study, the study treatment must be immediately discontinued. Pregnancy information for a female patient should be reported **within 24 hours** from the time the investigator first becomes aware of a pregnancy or its outcome. This should be performed by completing a Pregnancy Form and faxing it to Taiho Pharmacovigilance or designee.

New and/or corrected information regarding the pregnancy obtained after submitting the initial Pregnancy Form must be submitted by faxing an updated Pregnancy Form to Taiho Pharmacovigilance or designee.

If outcome of the pregnancy is a stillbirth, congenital anomaly/birth defect, or a serious event in the mother, report as an SAE to Taiho Pharmacovigilance or designee.

#### 10.84 Medication Errors

A **medication error** is defined as any accidental incorrect administration of a medicinal product. The error may be related to the administration of a wrong medication, nature of the medication, route of administration, dosage or frequency of the treatment as specified in this protocol (including omission of one or more administrations).

- Medication errors with study drugs and concomitant medication treatment will not be reported unless they result in an AE.
- Medication errors with study drugs that result in an overdose will be reported as an AE.
- Medication errors with study drugs that do not result in an AE should be handled as follows:
  - If it results in the omission of an administration, an incorrect dose (relative to that specified in this protocol), or the administration of more than the prescribed dose (but does not meet the overdose criteria), it will be identified through the recording of study drug accountability data in the CRF and does not need to be reported as an AE.
  - If it results in an overdose, incorrect route of administration, or administration of an incorrect study drug, it will be reported as an AE.

Based on the above criteria, medication errors that are captured as an AE on the CRF should be reported to Taiho Pharmacovigilance or designee within 24 hours from the time the investigator first becomes aware of its occurrence following the same process as described for the SAEs even if it does not meet any of the criteria of an SAE.

## 10.85 Overdose

An overdose with trifluridine/tipiracil for this clinical trial is defined as:

• Taking a dose beyond the recommended dose in 1 day or beyond the recommended total dose in each cycle.

An accidental or intentional overdose with trifluridine/tipiracil regardless of whether it is associated with an AE (even if not fulfilling a seriousness criterion) is to be captured as an AE on the CRF and reported to Taiho Pharmacovigilance or designee within 24 hours from the time the investigator first becomes aware of its occurrence following the same process as described for the SAEs.

There is no known antidote available in case of trifluridine/tipiracil overdose. Overdose should be managed aggressively with close monitoring and administration of prophylactic and symptomatic therapies to prevent or correct potential side effects.

An accidental or intentional overdose for concomitant medication should only be reported if it is associated with an AE.

To Report to Taiho Pharmacovigilance:

Protocol Version Date: 14Apr2020

#### 11.0 **Treatment Evaluation/Measurement of Effect**

NOTE: This study uses protocol RECIST v1.1 template dated 2/16/2011. See the footnote for the table regarding measurable disease in Section 11.44, as it pertains to data collection and analysis.

Response and progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guidelines (version 1.1) (Eisenhauer et al)<sup>13</sup>. Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the short axis measurements in the case of lymph nodes are used in the RECIST guideline.

#### Schedule of Evaluations 11.1

For the purposes of this study, patients should be reevaluated every 8 weeks. In addition to a baseline scan, confirmatory scans should also be obtained 8 weeks following initial documentation of objective response.

#### Definitions of Measurable and Non-Measurable Disease 11.2

#### 11.21 Measurable Disease

- A non-nodal lesion is considered measurable if its longest diameter can be accurately measured as  $\ge 2.0$  cm with chest x-ray, or as  $\ge 1.0$  cm with CT scan, CT component of a PET/CT, or MRI.
- 11.212 A superficial non-nodal lesion is measurable if its longest diameter is ≥1.0 cm in diameter as assessed using calipers (e.g. skin nodules) or imaging. In the case of skin lesions, documentation by color photography, including a ruler to estimate the size of the lesion, is recommended.
- A malignant lymph node is considered measurable if its short axis is 11.213 >1.5 cm when assessed by CT scan (CT scan slice thickness recommended to be no greater than 5 mm).

NOTE: Tumor lesions in a previously irradiated area are considered measurable disease under the following conditions:

- a) New lesion that has developed after radiation is completed
- b) Definite increase in the size of the previously irradiated lesion.

#### 11.22 Non-Measurable Disease

All other lesions (or sites of disease) are considered non-measurable disease, including pathological nodes (those with a short axis  $\geq 1.0$  to < 1.5 cm). Bone lesions, leptomeningeal disease, ascites, pleural/pericardial effusions, lymphangitis cutis/pulmonis, inflammatory breast disease, and abdominal masses (not followed by CT or MRI), are considered as non-measurable as well.

Note: 'Cystic lesions' thought to represent cystic metastases can be considered as measurable lesions, if they meet the definition of measurability described above. However, if non-cystic lesions are present in the same patient, these are preferred for selection as target lesions. In addition, lymph nodes that have a short axis < 1.0 cm are considered non- pathological (i.e., normal) and should not be recorded or followed.

<sup>&</sup>lt;sup>13</sup> Eisenhauer EA, Therasse P, Bogaert J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumors: revised RECIST guideline (version 1.1). Eur J Cancer 45(2): 228-247, 2009.

## 11.3 Guidelines for Evaluation of Measurable Disease

#### 11.31 Measurement Methods:

- All measurements should be recorded in metric notation (i.e., decimal fractions of centimeters) using a ruler or calipers.
- The same method of assessment and the same technique must be used to characterize each identified and reported lesion at baseline and during follow-up. For patients having only lesions measuring at least 1 cm to less than 2 cm must use CT imaging for both pre- and post-treatment tumor assessments.
- Imaging-based evaluation is preferred to evaluation by clinical examination when both methods have been used at the same evaluation to assess the antitumor effect of a treatment.

## 11.32 Acceptable Modalities for Measurable Disease:

Conventional CT and MRI: This guideline has defined measurability of lesions on CT scan based on the assumption that CT slice thickness is 5 mm or less. If CT scans have slice thickness greater than 5 mm, the minimum size for a measurable lesion should be twice the slice thickness.

- As with CT, if an MRI is performed, the technical specifications of the scanning sequences used should be optimized for the evaluation of the type and site of disease. The lesions should be measured on the same pulse sequence. Ideally, the same type of scanner should be used and the image acquisition protocol should be followed as closely as possible to prior scans. Body scans should be performed with breath-hold scanning techniques, if possible.
- PET-CT: If the site can document that the CT performed as part of a PET-CT is of identical diagnostic quality to a diagnostic CT (with IV and oral contrast), then the CT portion of the PET-CT can be used for RECIST measurements and can be used interchangeably with conventional CT in accurately measuring cancer lesions over time.
- Chest X-ray: Lesions on chest x-ray are acceptable as measurable lesions when they are clearly defined and surrounded by aerated lung. However, CT scans are preferable.
- Physical Examination: For superficial non-nodal lesions, physical examination is acceptable, but imaging is preferable, if both can be done. In the case of skin lesions, documentation by color photography, including a ruler to estimate the size of the lesion, is recommended.
- FDG-PET: FDG-PET scanning is allowed to complement CT scanning in assessment of progressive disease [PD] and particularly possible 'new' disease. A 'positive' FDG-PET scanned lesion is defined as one which is FDG avid with an update greater than twice that of the surrounding tissue on the attenuation corrected image; otherwise, an FDG-PET scanned lesion is considered 'negative.' New lesions on the basis of FDG-PET imaging can be identified according to the following algorithm:
  - a. Negative FDG-PET at baseline with a positive FDG-PET at follow-up is a sign of PD based on a new lesion.
  - b. No FDG-PET at baseline and a positive FDG-PET at follow-up:

- i. If the positive FDG-PET at follow-up corresponds to a new site of disease confirmed by CT, this is PD.
- ii. If the positive FDG-PET at follow-up is not confirmed as a new site of disease on CT at the same evaluation, additional follow-up CT scans (i.e., additional follow-up scans at least 4 weeks later) are needed to determine if there is truly progression occurring at that site. In this situation, the date of PD will be the date of the initial abnormal PDG-PET scan.
- iii. If the positive FDG-PET at follow-up corresponds to a pre-existing site of disease on CT that is not progressing.

## 11.33 Measurement at Follow-up Evaluation:

A subsequent scan must be obtained 8 weeks following initial documentation of an objective status of either complete response (CR) or partial response (PR). In the case of stable disease (SD), follow-up measurements must have met the SD criteria at least once after study entry at a minimum interval of 8 weeks (see Section 11.44).

The cytological confirmation of the neoplastic origin of any effusion that appears or worsens during treatment when the measurable tumor has met criteria for response or stable disease is mandatory to differentiate between response or stable disease (an effusion may be a side effect of the treatment) and progressive disease.

• Cytologic and histologic techniques can be used to differentiate between PR and CR in rare cases (e.g., residual lesions in tumor types such as germ cell tumors, where known residual benign tumors can remain.)

## 11.4 Measurement of Effect

#### 11.41 Target Lesions & Target Lymph Nodes

- Measurable lesions (as defined in Section 11.21) up to a maximum of 5 lesions representative of all involved organs, should be identified as "Target Lesions" and recorded and measured at baseline. These lesions can be non-nodal or nodal (as defined in 11.21), where no more than 2 lesions are from the same organ and no more than 2 malignant nodal lesions are selected.
   Note: If fewer than 5 target lesions and target lymph nodes are identified (as there often will be), there is no reason to perform additional studies beyond those specified in the protocol to discover new lesions.
- Target lesions and target lymph nodes should be selected on the basis of their size, be representative of all involved sites of disease, but in addition should be those that lend themselves to reproducible repeated measurements. It may be the case that, on occasion, the largest lesion (or malignant lymph node) does not lend itself to reproducible measurements in which circumstance the next largest lesion (or malignant lymph node) which can be measured reproducibly should be selected.
- Baseline Sum of Dimensions (BSD): A sum of the longest diameter for all target lesions plus the sum of the short axis of all the target lymph nodes will be calculated and reported as the baseline sum of dimensions (BSD). The
BSD will be used as reference to further characterize any objective tumor response in the measurable dimension of the disease.

- Post-Baseline Sum of the Dimensions (PBSD): A sum of the longest diameter for all target lesions plus the sum of the short axis of all the target lymph nodes will be calculated and reported as the post-baseline sum of dimensions (PBSD). If the radiologist is able to provide an actual measure for the target lesion (or target lymph node), that should be recorded, even if it is below 0.5 cm. If the target lesion (or target lymph node) is believed to be present and is faintly seen but too small to measure, a default value of 0.5 cm should be assigned. If it is the opinion of the radiologist that the target lesion or target lymph node has likely disappeared, the measurement should be recorded as 0 cm.
- The minimum sum of the dimensions (MSD) is the minimum of the BSD and the PBSD.

## 11.42 Non-Target Lesions & Non-Target Lymph Nodes

Non-measurable sites of disease (Section 11.22) are classified as non-target lesions or non-target lymph nodes and should also be recorded at baseline. These lesions and lymph nodes should be followed in accord with 11.433.

#### 11.43 Response Criteria

#### 11.431 Measurement

All target lesions and target lymph nodes followed by CT/MRI/PET-CT/Chest X-ray/physical examination must be measured on re-evaluation at evaluation times specified in Section 11.1. Specifically, a change in objective status to either a PR or CR cannot be done without re-measuring target lesions and target lymph nodes.

**Note:** Non-target lesions and non-target lymph nodes should be evaluated at each assessment, especially in the case of first response or confirmation of response. In selected circumstances, certain non-target organs may be evaluated less frequently. For example, bone scans may need to be repeated only when complete response is identified in target disease or when progression in bone is suspected.

#### 11.432 Evaluation of Target Lesions

**Complete Response (CR)**: All of the following must be true:

- a. Disappearance of all target lesions.
- b. Each target lymph node must have reduction in short axis to <1.0 cm.

Partial Response (PR): At least a 30% decrease in PBSD (sum of the longest diameter for all target lesions plus the sum of the short axis of all the target lymph nodes at current evaluation) taking as reference the BSD (see Section 11.41).

**Progression (PD)**: At least one of the following must be true:

a. At least one new malignant lesion, which also includes any lymph node that was normal at baseline (<1.0 cm short axis) and increased to ≥1.0 cm short axis during follow-up.

- b. At least a 20% increase in PBSD (sum of the longest diameter for all target lesions plus the sum of the short axis of all the target lymph nodes at current evaluation) taking as reference the MSD (Section 11.41). In addition, the PBSD must also demonstrate an absolute increase of at least 0.5 cm from the MSD.
- c. See Section 11.32 for details in regards to the requirements for PD via FDG-PET imaging.

**Stable Disease (SD)**: Neither sufficient shrinkage to qualify for PR, nor sufficient increase to qualify for PD taking as reference the MSD.

## 11.433 Evaluation of Non-Target Lesions & Non-target Lymph Nodes

Complete Response (CR): All of the following must be true:

- a. Disappearance of all non-target lesions.
- b. Each non-target lymph node must have a reduction in short axis to <1.0 cm.

**Non-CR/Non-PD**: Persistence of one or more non-target lesions or non-target lymph nodes.

**Progression (PD)**: At least one of the following must be true:

- a. At least one new malignant lesion, which also includes any lymph node that was normal at baseline (<1.0 cm short axis) and increased to ≥1.0 cm short axis during follow-up.
- b. Unequivocal progression of existing non-target lesions and non-target lymph nodes. (NOTE: Unequivocal progression should not normally trump target lesion and target lymph node status. It must be representative of overall disease status change.)
- c. See Section 11.32 for details in regards to the requirements for PD via FDG-PET imaging.

## 11.44 Overall Objective Status

The overall objective status for an evaluation is determined by combining the patient's status on target lesions, target lymph nodes, non-target lesions, non-target lymph nodes, and new disease as defined in the following tables:

#### 11.441 For Patients with Measurable Disease

| | Non-Target Lesions & | | |
|---|---|---|---|
| Target Lesions & | Non-Target Lymph | New | Overall Objective |
| Target Lymph Nodes | Nodes | Sites of Disease | Status |
| CR | CR | No | CR |
| CR | Non-CR/Non-PD | No | PR |
| PR | CR | No | PR |
| FK | Non-CR/Non-PD | INO | ΓK |
| CR/PR | Not All Evaluated* | No | PR** |
| | CR | | |
| SD | Non-CR/Non-PD | No | SD |
| | Not All Evaluated* | | |

| Target Lesions &<br>Target Lymph Nodes | Non-Target Lesions &<br>Non-Target Lymph<br>Nodes | New<br>Sites of Disease | Overall Objective<br>Status |
|---|---|---|---|
| Not all evaluated | CR<br>Non-CR/Non-PD<br>Not All Evaluated* | No | Not Evaluated (NE) |
| PD | Unequivocal PD<br>CR<br>Non-CR/Non-PD<br>Not All Evaluated* | Yes or No | PD |
| CR/PR/SD/PD/Not all<br>Evaluated | Unequivocal PD | Yes or No | PD |
| CR/PR/SD/PD/Not all<br>Evaluated | CR<br>Non-CR/Non-PD<br>Not All Evaluated* | Yes | PD |

<sup>\*</sup>See Section 11.431

## 11.45 Symptomatic Deterioration

Patients with global deterioration of health status requiring discontinuation of treatment without objective evidence of disease progression at that time, and not either related to study treatment or other medical conditions, should be reported as PD due to "symptomatic deterioration." Every effort should be made to document the objective progression even after discontinuation of treatment due to symptomatic deterioration. A patient is classified as having PD due to "symptomatic deterioration" if any of the following occur that are not either related to study treatment or other medical conditions:

- Weight loss >10% of body weight.
- Worsening of tumor-related symptoms.
- Decline in performance status of >1 level on ECOG scale.

#### 12.0 Descriptive Factors

- 12.1 Prior treatment: 1 vs 2 vs 3+
- 12.2 Primary site of tumor: Gallbladder vs intrahepatic vs extrahepatic biliary tract cancer
- 12.3 Degree of differentiation: Well vs moderately vs poorly differentiated vs undifferentiated/anaplastic vs cannot be assessed/unknown
- 12.4 ECOG performance status: 0 vs 1
- 12.5 Prior treatment with fluoropyrimidine based regimen: Yes vs no

## 13.0 Treatment/Follow-up Decision at Evaluation of Patient

#### 13.1 Continuation of treatment

Patients who are CR, PR, or SD will continue treatment per protocol.

<sup>\*\*</sup> NOTE: This study uses the protocol RECIST v1.1 template dated 2/16/2011. For data collection and analysis purposes the objective status changed from SD to PR in the MCCC protocol RECIST v1.1 template as of 2/16/2011 and to match RECIST v1.1 requirement.

## 13.2 Progressive disease (PD)

Patients who develop PD while receiving therapy will go to the event-monitoring phase.

## 13.3 Off protocol treatment

Patients who go off protocol treatment for reasons other than PD will go to the event-monitoring phase per Section 4.0. Treatment decision during event-monitoring phase is at the discretion of the treating physician.

## 13.4 Duration of therapy for CR, PR or SD

Patients who achieve a CR, PR or SD will continue to receive treatment per protocol until they develop PD or unacceptable toxicity.

## 13.5 Definition of Ineligible

A patient is deemed ineligible if after registration, it is determined that at the time of registration, the patient did not satisfy each and every eligibility criteria for study entry. The patient may continue treatment off-protocol at the discretion of the physician as long as there are no safety concerns, and the patient was properly registered. The patient will go directly to the event-monitoring phase of the study (or off study, if applicable).

- If the patient received treatment, all data up until the point of confirmation of ineligibility must be submitted. Event monitoring will be required per Section 18.0 of the protocol.
- If the patient never received treatment, on-study material must be submitted. Event monitoring will be required per Section 4.0 of the protocol.

## 13.6 Definition of Major Violation

A patient is deemed a major violation, if protocol requirements regarding treatment in cycle 1 of the initial therapy are severely violated that evaluability for primary end point is questionable. All data up until the point of confirmation of a major violation must be submitted. The patient will go directly to the event-monitoring phase of the study. The patient may continue treatment off-protocol at the discretion of the physician as long as there are no safety concerns, and the patient was properly registered. Event monitoring will be required per Section 4.0 of the protocol.

#### 13.7 Definition of Cancel

A patient is deemed a *cancel* if he/she is removed from the study for any reason before any study treatment is given. On-study material and the End of Active Treatment/Cancel Notification Form must be submitted. No further data submission is necessary.

#### 13.8 Patient removal from study

Patients may be removed from treatment on this study for any of the following reasons:

- Progression of disease
- Noncompliance with study procedures
- Patient's request to withdraw from the study or refusal of further therapy
- Unacceptable adverse events: A patient may be removed from the study for any complication of treatment that the investigator feels is life threatening
- Investigator discretion
- Dose delay >28 days for treatment related AE NOTE: If a patient has clinical benefit from the study treatment, patient may continue on study at investigator discretion

## 14.0 Body Fluid Biospecimens

## 14.1 Summary Table of Research Blood and Body Fluid Specimens to be Collected for this Protocol

| Research (Section for more information) | Specimen Purpose (check all that apply) | Mandatory<br>or Optional | Blood or<br>Body Fluid<br>being<br>Collected | Type of<br>Collection<br>Tube (color<br>of tube top) | Volume to<br>collect per<br>tube (# of<br>tubes to be<br>collected) | Baseline<br>prior to<br>Cycle 1,<br>Day 1 | Cycle 3,<br>Day 1 | End of<br>treatment | Process<br>at site?<br>(Yes or<br>No) | Temperature<br>Conditions<br>for Storage<br>/Shipping |
|---|---|---|---|---|---|---|---|---|---|---|
| Circulating biomarker<br>work<br>(Section 14.2 and 14.3) | ☐ Correlative ☐ Eligibility Confirmation ☐ Banking ☐ Other (specify) | Mandatory | Whole blood<br>for DNA,<br>buffy coat,<br>WBCs and<br>plasma* | EDTA tube (purple top) | 10 mL<br>(1) | X | X | X | Yes | Frozen on dry ice |
| cfDNA based studies<br>(Section 14.2 and 14.3) | ☐ Correlative ☐ Eligibility Confirmation ☐ Banking ☐ Other (specify) | Mandatory | Whole blood<br>for platelet<br>poor plasma | Streck<br>cfDNA BCT | 10 mL<br>(2) | X | X | X | None | Ship same day<br>at ambient<br>temperature |
| CTC based studies (Section 14.2 and 14.3) | ☐ Correlative ☐ Eligibility Confirmation ☐ Banking ☐ Other (specify) | Mandatory | Whole blood<br>for CTCs | AccuCyte<br>tube | 10 mL<br>(1) | X | X | X | None | Ship same day<br>at ambient<br>temperature |

<sup>\*</sup> DNA extraction from whole blood to be done at each site

## 14.2 Collection and Processing

- 14.21 Sample collection should be restricted to Monday Thursday. However, if the subject can only be seen on a Friday, please contact the Biospecimen Resource Manager for additional instructions (see protocol resource pages for contact information).
- 14.22 Specimen tube(s) must be labeled with the protocol number, study patient ID number, and the time and date of the blood draw.
- 14.23 Blood/blood products must be collected and shipped according to specific instructions provided in the kit and the table above.

## 14.3 Shipping

- 14.31 Verify that ALL sections of the Blood Specimen Submission Form (see Forms Packet), BAP Requisition Form (provided in kit), and specimen collection labels are completed and filled in correctly. Enter information from the Blood Specimen Submission Form into the remote data entry system within 7 days after specimen collection (see Forms Packet).
- 14.32 Specimens collected in the Streck cfDNA BCT and AccuCyte tubes should be shipped at ambient temperature on the same day they are drawn.
- 14.33 Specimens collected in EDTA tubes should be processed for DNA from whole blood, a buffy coat back up and plasma aliquots then stored frozen. NOTE: DNA extraction must be done at site where it's collected.
- 14.34 Samples should be shipped to BAP Freezer Mondays Thursdays according to kit instructions. Samples should not be sent on weekends or just prior to federal holidays. (If samples can only be shipped on Fridays, please contact the Biospecimen Resource Manager for additional instructions.)

## 14.4 Processing

NOTE: BAP Shared Resource will process the specimens.

- 14.41 Double spun, platelet poor plasma will be derived from the Streck cfDNA BCT tubes using established laboratory processes, and stored at ≤-65°C by BAP.
- 14.42 DNA will be extracted from whole blood, and white blood cells and plasma will be derived from remaining blood from the EDTA tubes, divided into aliquots, and stored at ≤-65°C by BAP according to patient consent information.
- Whole blood collected in the AccuCyte tubes will be provided directly to laboratory at Mayo Clinic Rochester to isolate and retain CTCs.
- 14.44 As part of ongoing research at the Mayo Clinic, we will retain residual whole blood, white blood cells, CTCs, DNA, and plasma for future research studies, according to patient consent information. Samples will be stored until specific analyses are identified and may be used for exploratory biomarker analyses, validation studies, or potential diagnostic development. As protocols are developed, they will be presented for IRB review and approval.

## 14.5 Background and Methodology

#### 14.51 ctDNA

Detection of cancer specific mutations from the peripheral blood is an area of active investigation in many different types of cancers. An accumulating body of literature confirms an excellent correlation between mutations found in cancer tissues and mutations detected in cfDNA from the same patients. (Kim et al. 2015) Changes in cfDNA also correlate well with tumor marker dynamics in serial sampling, suggesting that cfDNA mutant allele fraction changes reflect changes in disease burden over time and treatment. Plasma based DNA mutation detection should therefore provide longitudinal changes in the representative genomic landscape of the malignancy in a non-invasive manner, overcoming the two major limitations of tissue based DNA mutation analysis (invasiveness and limited sampling from a genetically heterogeneous tumor). (Diehl et al. 2005; Diehl et al. 2008; Dawson et al. 2013)

10 mL whole blood samples will be collected in Streck cfDNA BCT tubes. These specimens will be shipped immediately at ambient temperature to Mayo Clinic Rochester and then processed to aliquots of platelet poor plasma within 7 days of collection using standard protocols. Samples will be stored until we are ready for DNA extraction and mutational analysis.

Mutation analysis will be performed on the baseline cfDNA samples including FGFR and HER-2. Selected mutations identified at baseline will be verified and quantified in all cfDNA samples using ultrasensitive digital droplet PCR based assays.

## 14.52 CTCs

That CTCs have biologic relevance in epithelial malignancies is increasingly clear, as their relative abundance in the peripheral blood has strong correlations with disease related outcomes in early stage and advanced breast cancer. (Liu et al. 2009; Liu 2014) Beyond simple enumeration, molecular profiling of these cells may provide clinically relevant predictive information to guide the selection of therapy. Deriving detailed molecular signatures for isolated CTCs may also facilitate drug discovery by assessing the markers unique to progression, such that relapsing patients may be treated for their current molecular disease.

The RareCyte CTC technology is a comprehensive, reproducible and highly sensitive dual-platform for collecting, identifying and analyzing CTCs that does not rely on EpCAM expression for enrichment.6 The front end AccuCyte system is based fundamentally on the density of CTCs, which is within the range of the buffy coat; a unique separation tube and collector device allow for virtually complete harvesting of the buffy coat into a small volume for application to a microscopic slide without cell lysis or wash steps, a potential source of CTC loss. The follow-up CyteFinder system is an automated scanning digital microscope and image analysis system that presents high-resolution images of candidate cells stained with well-characterized markers before definitive classification as a CTC. Importantly, CyteFinder includes an integrated device (CytePicker<sup>TM</sup>) for CTC retrieval that is mechanically precise, enabling the isolation of DNA derived from single or pooled CTCs advanced genomic analyses including the detection of specific mutations and targeted NGS. The Mayo group has established

MC1941 44 MCCC Amendment 1

experience detecting and isolated purified CTCs from breast cancer patients, as well as the capability to design 4- or 6-marker panels to capture specific phenotypic populations of CTCs.

10 mL whole blood samples will be collected in AccuCyte Blood Collection Tubes, which contain the proprietary RareCyte cell preservative. These samples will be shipped immediately at ambient temperature to Mayo Clinic Rochester and then processed through the RareCyte system within 3 days of collection. CTCs will be captured onto glass slides (8 slides per blood sample) for subsequent immunofluorescent staining, selection, and single cell isolation. The markers used for CTC identification will include DAPI or SYTOX orange, cytokeratin, and EpCAM at a minimum. CD45 will be used to distinguish WBCs (CD45 positive) from CTCs (CD45 negative). Pure populations of CTCs will then be isolated and stored for subsequent molecular analyses, as yet to be determined.

MC1941 45 MCCC Amendment 1

## 15.0 Drug Information

## **15.1** Trifluridine/tipiracil (FTD/TPI, TAS-102, Lonsurf®)

## 15.11 Background

Trifluridine/tipiracil (FTD/TPI) is an orally available combination drug of an antineoplastic thymidine-based nucleoside analogue, 1M trifluridine, and 0.5 M tipiracil hydrochloride. Trifluridine is incorporated into deoxyribonucleic acid of tumor cells following phosphorylation. Tipiracil inhibits degradation of trifluridine by thymidine phosphorylase.

#### 15.12 Formulation

Trifluridine/tipiracil contains trifluridine (FTD) and tipiracil (TPI) as active ingredients with a molar ratio of 1:0.5. Trifluridine/tipiracil drug products are immediate-released film coated tablets, with two strengths of 15 mg and 20 mg (expressed as trifluridine). The inactive ingredients of the FTD/TPII 15 mg and 20 mg tablets are lactose monohydrate, pregelatinized starch, stearic acid, hypromellose, polyethylene glycol, titanium dioxide, red ferric oxide (only 20 mg tablet), and magnesium stearate.

Trifluridine/tipiracil (FTD/TPI) tablet (15 mg) contains 15 mg trifluridine and 7.065 mg tipiracil as active ingredients. The appearance is white, round, biconvex, film-coated, tablets.

Trifluridine/tipiracil (FTD/TPI) tablet (20 mg) contains 20 mg trifluridine and 9.42 mg tipiracil as active ingredients. The appearance is pale red, round, biconvex, film-coated,tablet.

## 15.13 Preparation and storage

Store at 20°C to 25°C (68°F to 77°F); excursions are permitted from 15°C to 30°C (59°F to 86°F). If stored outside of original bottle, discard after 30 days.

## 15.14 Administration

Please see Pharmacy Manual provided by Taiho Oncology for this study. Recommended to take within 1 hour after completion of the morning and evening meals.

The recommended dosage of FTD/TPI is 35 mg/m² up to a maximum of 80 mg per dose (based on the trifluridine component) orally twice daily with food on Days 1 through 5 and Days 8 through 12 of each 28-day cycle until disease progression or unacceptable toxicity. Round dose to the nearest 5 mg increment. Instruct patients to swallow FTD/TPI tablets whole.

Instruct patients not to retake doses of FTD/TPI that are vomited or missed and to continue with the next scheduled dose.

#### 15.15 Pharmacokinetic information

Protein Binding: Trifluridine: >96% (primarily to albumin); Tipiracil: <8%

Metabolism: Trifluridine and tipiracil are not metabolized by cytochrome P450 (CYP) enzymes. Trifluridine is mainly eliminated by metabolism via thymidine phosphorylase to form an inactive metabolite, 5-(trifluoromethyl) uracil (FTY) Half-life elimination: Trifluridine: 2.1 hours (at steady state); Tipiracil: 2.4 hours (at steady state)

Time to peak, plasma: ~2 hours

Excretion: Trifluridine: Urine (55% [as inactive metabolite FTY and trifluridine glucuronide isomers]; <3% [as unchanged drug]; feces (<3% [as unchanged drug]); expired air (<3%)

Tipiracil: Urine (~27% [as tipiracil and 6-HMU]; feces (50% [as tipiracil and 6-HMU])

## 15.16 Potential drug interactions

Caution is required when using drugs that are human thymidine kinase substrates, e.g., zidovudine. Such drugs, if used concomitantly with FTD/TPI, may theoretically compete with the effector of FTD/TPI, i.e., FTD, for activation via thymidine kinases. Therefore, when using antiviral drugs that are human thymidine kinase substrates, monitor for possible decreased efficacy of the antiviral agent, and consider switching to an alternative antiviral agent that is not a human thymidine kinase substrate such as: lamivudine, zalcitabine, didanosine, abacavir, etc.

#### 15.17 Known potential adverse events

## Very common known potential adverse events, ≥10%:

Blood and lymphatic: Anemia, leukopenia, neutropenia, thrombocytopenia

Gastrointestinal: Diarrhea, nausea, vomiting

General: Fatigue

Metabolism and nutrition: Decreased appetite

#### Common known potential adverse events, ≥1% - <10%

Blood and lymphatic: Febrile neutropenia, lymphopenia, monocytosis

Dermatologic: Alopecia, dry skin, Palmar-plantar erythrodysesthesia syndrome,

pruritis, rash

Gastrointestinal: Abdominal pain, constipation, oral disorder, stomatitis

General: Malaise, mucosal inflammation, edema, pyrexia

Hepatobiliary: Hyperbilirubinemia

Infections: Lower respiratory tract infection, upper respiratory tract infection Investigations: Blood alkaline phosphatase increased, hepatic enzyme increased,

weight decreased

Metabolism and nutrition: Hypoalbuminemia

Nervous System: Dizziness, dysgeusia, headache, peripheral neuropathy

Psychiatric: Insomnia

Renal and urinary: Proteinuria Respiratory: Cough, dyspnea

Vascular: Flushing

# Uncommon known potential adverse events, <1% (Limited to important or life-threatening):

Blood and lymphatic: Pancytopenia

Gastrointestinal: Ascites, colitis, ileus, acute pancreatitis, subileus

General: General physical health deterioration

Infections: Bacterial infection, biliary tract infection, enteritis infection, urinary

tract infection

Investigations: Blood lactate dehydrogenase increased

Metabolism and nutrition: Dehydration Respiratory: Pulmonary embolism

## 15.18 Drug procurement

FTD/TPI will be provided free of charge by Taiho Oncology.

## 15.19 Nursing guidelines

- 15.191 Instruct Patients to take FTD/TPI within 1 hour after completion of morning or evening meal with a glass of water.
- 15.192 Patients may experience fatigue. Instruct patients in energy conserving lifestyle.
- 15.193 GI side effects are common, including nausea, decreased appetite, diarrhea, vomiting, and abdominal pain.
- 15.194 Cytopenias are common. Monitor CBC w/diff and instruct patients to report any signs or symptoms of infection and/or unusual bruising or bleeding to the study team.
- 15.195 Rarely Pulmonary embolism has been reported with this agent. Instruct patient to report any shortness of breath or chest pain to study team and/or seek out emergency medical attention.
- 15.196 Although uncommon, warn patients of the possibility of alopecia.

## 15.2 Irinotecan (Camptosar®, CPT11)

## 15.21 Background

Irinotecan and its active metabolite SN-38 bind to the topoisomerase I-DNA complex and prevent religation of the cleaved DNA strand. This results in the accumulation of cleavable complexes and double-strand DNA breaks. As mammalian cells cannot efficiently repair these breaks, cell death consistent with S-phase cell cycle specificity occurs, leading to termination of cellular replication.

#### 15.22 Formulation

Commercially available for injection 20 mg/mL (2 mL, 5 mL, 25 mL) [contains sorbitol 45 mg/mL; do not use in patients with hereditary fructose intolerance]..

#### 15.23 Preparation and storage

Store intact vials at controlled room temperature 15-30°C (59-86°F) and protect from light. Doses should be diluted in 250-500 mL  $D_5W$  or 0.9% NaCl to a final concentration of 0.12-2.8 mg/mL. Solutions diluted in D5W are stable for 24 hours at room temperature or 48 hours under refrigeration at 2°C to 8°C. Solutions diluted in 0.9% NaCl may precipitate if refrigerated. Do not freeze.

#### 15.24 Administration

Administer as IV infusion, usually over 90 minutes.

#### 15.25 Pharmacokinetic information

Distribution: V<sub>d</sub>: 33-150 L/m<sup>2</sup>

Protein binding, plasma: Predominantly albumin; Parent drug: 30% to 68%, SN-38 (active metabolite): ~95%

Metabolism: Primarily hepatic to SN-38 (active metabolite) by carboxylesterase enzymes; SN-38 undergoes conjugation by UDP- glucuronosyl transferase 1A1 (UGT1A1) to form a glucuronide metabolite. Conversion of Irinotecan to SN-38 is decreased and glucoronidation of SN-38 is increased in patients who smoke cigarettes, resulting in lower levels of the metabolite and overall decreased systemic exposure. SN-38 is increased by UGT1A1\*28 polymorphism (10% of North Americans are homozygous for UGT1A1\*28 allele). Patients homozygous for the UGT1A1\*28 allele are at increased risk of neutropenia; initial one-level dose reduction should be considered for both single-agent and combination regimens. The lactones of both Irinotecan and SN-38 undergo hydrolysis to inactive hydroxyl acid forms.

Half-life elimination: SN-38: mean terminal 10-20 hours

Time to peak: SN-38: Following 90-minute infusion  $\sim$ 1 hour

Excretion: Within 24 hours: urine: Irinotecan (11% to 20%), metabolites (SN-38

<1%, SN-38 glucuronide, 3%)

## 15.26 Potential drug interactions

Cytochrome P450 Effect: Substrate (major) of CYP2B6, 3A4, P-glycoprotein, SLCO1B1 and UGT1A1

Increased Effect/Toxicity: CYP2B6 and CYP3A4 inhibitors may increase the levels/effects of irinotecan. Bevacizumab may increase the adverse effects of Irinotecan (e.g., diarrhea, neutropenia). Ketoconazole increases the levels/effects of irinotecan and active metabolite; discontinue ketoconazole 1 week prior to irinotecan therapy; concurrent use is contraindicated.

**Decreased Effect:** CYP2B6 and CYP3A4 inducers may decrease the levels/effects of irinotecan.

**Ethanol/Nutrition/Herb Interactions** Herb/Nutraceutical: St John's wort decreases therapeutic effect of irinotecan; discontinue ≥2weeks prior to irinotecan therapy; concurrent use is contraindicated.

## 15.27 Known potential adverse events

Consult the package insert for the most current and complete information including U.S. Boxed Warnings pertaining to severe diarrhea and severe myelosuppression.

#### Common known potential adverse events, >10%:

Cardiovascular: Vasodilation

Central nervous system: Cholinergic toxicity (includes rhinitis, increased salivation, miosis, lacrimation, diaphoresis, flushing and intestinal hyperperistalsis); fever, pain, dizziness, insomnia, headache, chills

Dermatologic: Alopecia, rash

Endocrine & metabolic: Dehydration

Gastrointestinal: Late onset diarrhea, early onset diarrhea, nausea, abdominal pain, vomiting, cramps, anorexia, constipation, mucositis, weight loss, flatulence, stomatitis

Hematologic: Anemia, leukopenia, thrombocytopenia, neutropenia

Hepatic: Bilirubin increased, alkaline phosphatase increased

Neuromuscular & skeletal: Weakness, back pain

Respiratory: Dyspnea, cough, rhinitis Miscellaneous: Diaphoresis, infection

#### Less common known adverse events, 1% - 10%:

Cardiovascular: Edema, hypotension, thromboembolic events

Central nervous system: Somnolence, confusion Gastrointestinal: Abdominal fullness, dyspepsia

Hematologic: Neutropenic fever, hemorrhage, neutropenic infection

Hepatic: AST increased, ascites and/or jaundice

Respiratory: Pneumonia

# Rare known potential adverse events, <1% (Limited to important or life-threatening):

ALT increased, amylase increased, anaphylactoid reaction, anaphylaxis, angina, arterial thrombosis, bleeding, bradycardia, cardiac arrest, cerebral infarct, cerebrovascular accident, circulatory failure, colitis, dysrhythmia, embolus, gastrointestinal bleeding, gastrointestinal obstruction, hepatomegaly, hyperglycemia, hypersensitivity, hyponatremia, ileus, interstitial pulmonary disease (IPD), intestinal perforation, ischemic colitis, lipase increased, lymphocytopenia, megacolon, MI, myocardial ischemia, neutropenic typhlitis, pancreatitis, paresthesia, peripheral vascular disorder, pulmonary embolus, pulmonary toxicity (dyspnea, fever, reticulonodular infiltrates on chest x-ray), renal failure (acute), renal impairment, syncope, thrombophlebitis, thrombosis, typhlitis, ulceration, ulcerative colitis

#### 15.28 Drug procurement

Commercial supplies. Pharmacies or clinics shall obtain supplies from normal commercial supply chain or wholesaler.

## 15.29 Nursing guidelines

- 15.291 If possible, check for any history of hypersensitivity reaction to any previous drug formulated with polysorbate 80.
- 15.292 Cholinergic symptoms of lacrimation, nasal congestion, diaphoresis, flushing, ABD cramping, and diarrhea can occur at the beginning, during, or immediately after the CPT-11 infusion. It is suggested that the patient remain in the treatment area for a minimum of one hour following the completion of the <u>very first CPT-11</u> infusion. If diarrhea occurs within one hour of infusion, refer to Section 9.2 for management.
- 15.293 Patient education is extremely important. Impress on the patient the importance of compliance with treatment of diarrhea management (see Section 9.1). Stress the need for prompt recognition and early intervention. Motivate the patient to report any complications

- immediately. The cholera-like syndrome can be unresponsive to conventional antidiarrheals and can result in severe dehydration.
- 15.294 Ondansetron and diphenhydramine should provide good relief from the nausea/vomiting/cramping. Avoid prochlorperazine on the day of treatment due to its association with akathisia (motor restlessness). Prochlorperazine may be taken between treatments.
- 15.295 Advise avoidance of excess caffeine, a GI stimulant. Avoid magnesium based antacids such as Mylanta, Maalox, Rolaids, MOM, Mag-Ox 400, and Tylenol with antacid.
- 15.296 The pulmonary toxicity seen is usually manifested by dyspnea beginning 42-175 days after treatment and occurs at a cumulative dose ranging from 400-1000 mg/m² (median 750). Instruct patient to report any cough or SOB.
- 15.297 Patients are at risk for developing eosinophilia and will improve on steroid therapy.
- 15.298 Hepatic enzyme elevations have been transient and did not require intervention.
- 15.299a Monitor CBC closely. Leukopenia occurs primarily as neutropenia but can be severe and dose-limiting. The simultaneous occurrence of Grade 4 diarrhea and Grade 4 neutropenia are rare but may render the patient more susceptible to polymicrobial sepsis and potentially death.
- 15.299b Advise patients of probable hair loss.

## 16.0 Statistical Considerations and Methodology

#### 16.1 Overview

This protocol will assess the efficacy of trifluridine/tipiracil plus irinotecan in patients with refractory cholangiocarcinoma using a two stage phase II study design. This single arm Phase II trial will assess the 16-week progression-free survival rate (by RECIST v1.1) associated with trifluridine/tipiracil plus irinotecan in patients with refractory cholangiocarcinoma. We will adopt a PFS rate of 10% as the null hypothesis and PFS rate of 30% as the alternative hypothesis. In addition to response, this study will also evaluate the overall response rate (ORR), progression-free survival (PFS), overall survival (OS), disease control rate (DCR), and adverse events.

## 16.11 Primary Endpoint

The primary endpoint for this study is 16-week progression-free survival associated with trifluridine/tipiracil plus irinotecan in patients with refractory cholangiocarcinoma.

## 16.2 Statistical Design

#### 16.21 Decision Rule

The largest success proportion where the proposed treatment regimen would be considered ineffective in this population is 10%, and the smallest success proportion that would warrant subsequent studies with the proposed regimen in this patient population is 30%. The following two stage design (Simon) uses 15 or 25 patients to test the null hypothesis that the true success proportion in a given patient population is at most 10%.

NOTE: We consider a success to be alive and progression-free by 16 weeks post-registration (i.e. stable disease, partial response, or complete response).

- 16.211 STAGE 1: Enter 15 patients into the study. If 1 or fewer successes are observed in the first 15 evaluable patients, we will consider this regimen ineffective in this patient population and terminate this study. Otherwise, if the number of successes is at least 2, we will proceed to Stage 2.
- 16.212 STAGE 2: Enter an additional 10 patients into the study. If 5 or fewer successes are observed in the first 25 evaluable patients, we will consider this regimen ineffective in this patient population. If 6 or more successes are observed in the first 25 evaluable patients, we may recommend further testing of this regimen in subsequent studies in this population.
- 16.213 Over Accrual: If more than the target number of patients are accrued, the additional patients will not be used to evaluate the stopping rule or used in any decision-making process. Analyses involving over accrued patients are discussed in Section 16.34.
- 16.214 NOTE: We will not suspend accrual between stages to allow the first 15 patients to become evaluable, unless undue toxicity is observed.

## 16.22 Sample Size

The two-stage study design to be utilized is fully described in Section 16.21. A minimum of 15 and a maximum of 25 evaluable patients will be accrued onto this phase II study unless undue toxicity is encountered. We anticipate accruing an additional 3 patients to account for ineligibility, cancellation, major treatment violation, or other reasons. Maximum projected accrual is therefore 28 patients.

## 16.23 Accrual Time and Study Duration

The anticipated accrual rate is approximately 2 patients per month. Therefore, the accrual period for this phase II study is expected to be between 7.5 and 14 months, depending upon whether patients are accrued beyond the first stage. The final analysis can begin approximately 18 months after the trial begins, i.e. as soon as the last patient has been observed for 4 months.

## 16.24 Power and Significance Level

Assuming that the number of successes is binomially distributed, the significance level is 0.05 and the probability of declaring that this regimen warrants further studies (i.e. statistical power) under various success proportions and the probability of stopping accrual after the first stage can be tabulated as a function of the true success proportion as shown in the following table.

| If the true success proportion is | 0.10 | 0.15 | 0.20 | 0.25 | 0.30 |
|---|---|---|---|---|---|
| then the probability of declaring that the regimen warrants further studies is | 0.03 | 0.16 | 0.38 | 0.61 | 0.80 |
| and the probability of stopping at stage 1 is | 0.56 | 0.31 | 0.17 | 0.08 | 0.04 |

#### 16.25 Other Considerations

Adverse events, quality/duration of response, and patterns of treatment failure observed in this study, as well as scientific discoveries or changes in standard care will be taken into account in any decision to terminate the study.

## 16.3 Analysis Plan

The analysis for this trial will commence at planned time points (see 16.2) and at the time the patients have become evaluable for the primary endpoint. Such a decision will be made by the Statistician and Study Chair, in accord with CCS Standard Operating Procedures, availability of data for secondary endpoints (eg, laboratory correlates), and the level of data maturity. It is anticipated that the earliest date in which the results will be made available via manuscript, abstract, or presentation format is when patients have been on study for 16 weeks (i.e. received second scan).

## 16.31 Primary Endpoint

#### 16.311 Definition

The primary endpoint of this trial is the progression-free survival rate. This is defined as the proportion of evaluable patients who are progression-free (stable disease, partial response, complete response) at 16 weeks. All patients meeting the eligibility criteria who have signed a consent form, begun treatment, and undergone restaging scans (unless deemed to have clinical progression by investigator) will be considered evaluable for the primary endpoint.

#### 16.312 Estimation

The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Confidence intervals for the true success proportion will be calculated according to the approach of Clopper and Pearson.

#### 16.313 Over Accrual

If more than the target number of patients are accrued, the additional patients will not be used to evaluate the stopping rule or used in any decision-making processes; however, they will be included in final point estimates and confidence intervals as though they were accrued in the final stage.

## 16.32 Secondary Endpoints

The following endpoints will be evaluated: overall response rate, progression-free survival, overall survival, and adverse events. For efficacy outcomes, the same population defined in Section 16.311 will be used as the evaluable population. For adverse event outcomes, all consented patients eligible to begin treatment will be evaluated.

## 16.321 Overall Response Rate (ORR):

Overall response rate is defined as the proportion of patients who experience either a partial response or complete response as their best response. ORR will be reported descriptively and a 95% confidence interval will be reported.

## 16.322 Disease Control Rate (DCR):

Disease control rate is defined as the proportion of patients who experience a partial response, complete response, or have stable disease as their best response. DCR will be reported descriptively and a 95% confidence interval will be reported.

## 16.322 Progression-Free Survival (PFS):

Progression-free survival is defined as the time from study entry to the first of either disease progression or death from any cause, where disease progression will be determined based on RECIST 1.1 criteria. PFS will be estimated using the Kaplan-Meier method. The median PFS and 95% confidence interval will be reported. Patients will be censored at the last disease assessment date.

## 16.323 Overall Survival (OS):

Overall survival is defined as the time from study entry to death from any cause. OS will be estimated using the Kaplan-Meier method. The median OS and 95% confidence interval will be reported. Patients will be censored at the date patient was last known to be alive.

#### 16.324 Adverse events

The maximum grade for each type of adverse event by patient will be summarized by frequencies and percentages using NCI CTCAE version 5.0. We will also closely monitor adverse events throughout the study.

#### 16.33 Correlative Research

- 16.331 To determine if CTCs or cfDNA at baseline will correlate with prognosis or response to therapy.
- 16.332 To determine if change in CTCs or cfDNA will correlate with efficacy endpoints.
- 16.333 To determine if drug response from a parallel *ex vivo* trial using patient-derived tumor organoid correlates with clinical response to trifluridine/tipiracil plus irinotecan.
- 16.334 To evaluate the role of thymidine kinase 1 (TK1) in predicting the clinical benefit of trifluridine/tipiracil plus irinotecan and discover potential mechanisms of resistance using patient-derived tumor organoid and pre-treatment biopsy specimen.

## 16.34 Exploratory Analysis

To explore the population of patients that received prior treatment with 5-FU, patients within this cohort will be evaluated for endpoints that may include, but not be limited to: PFS, safety and tolerability, ORR, DCR, and OS.

## 16.4 Data & Safety Monitoring

#### 16.41 Review

The study chair(s) and the study statistician will review the study at least twice a year to identify accrual, adverse event, and any endpoint problems that might be developing. The Mayo Clinic Cancer Center (MCCC) Data Safety Monitoring Board (DSMB) is responsible for reviewing accrual and safety data for this trial at least twice a year, based on reports provided by the MCCC Statistical Office.

## 16.42 Adverse events stopping rules

The stopping rules specified below are based on the knowledge available at study development. We note that the Adverse Event Stopping Rule may be adjusted in the event of either (1) the study re-opening to accrual or (2) at any time during the conduct of the trial and in consideration of newly acquired information regarding the adverse event profile of the treatment(s) under investigation. The study team may choose to suspend accrual because of unexpected adverse event profiles that have not crossed the specified rule below.

Accrual will be temporarily suspended to this study if at any time we observe events considered at least possibly related to study treatment (i.e. an adverse event with attribute specified as "possible", "probable", or "definite") that satisfy either of the following:

- if 3 or more patients in the first 10 treated patients experience a Grade 4 or 5 adverse event at least possibly related to study treatment with the exception of transient laboratory events or cytopenias that resolve/improve within 7 days.
- if after the first 10 patients have been treated, 30% of all patients enrolled and treated experience a Grade 4 or 5 adverse event with the exception of transient laboratory events or cytopenias that resolve/improve within 7 days

We note that we will review Grade 4 and 5 adverse events deemed "unrelated" or "unlikely to be related", to verify their attribution and to monitor the emergence of a previously unrecognized treatment-related adverse event.

## 16.5 Subset Analyses for Minorities

#### 16.51 Study availability

This study will be available to all eligible patients, regardless of gender, race or ethnic origin.

## 16.52 Statistical analysis by subset

There is no information currently available regarding differential effects of this regimen in subsets defined by race, gender, or ethnicity, and there is no reason to expect such differences to exist. Therefore, although the planned analyses will look for differences in treatment effect based on racial groupings, the sample size is not increased in order to provide additional power for subset analyses.

#### 16.53 Regional population

The geographical region served by MCCC has a population which includes approximately 3% minorities. Expected sizes of racial by gender subsets are shown in the following table:

| Accrual Targets | | | |
|---|---|---|---|
| | Sex/Gender | | |
| Ethnic Category | Females | Males | Total |
| Hispanic or Latino | 1 | 1 | 2 |
| Not Hispanic or Latino | 13 | 13 | 26 |
| Ethnic Category: Total of all subjects | 14 | 14 | 28 |
| Racial Category | | | |
| American Indian or Alaskan Native | 0 | 0 | 0 |
| Asian | 0 | 0 | 0 |
| Black or African American | 1 | 1 | 2 |
| Native Hawaiian or other Pacific Islander | 0 | 0 | 0 |
| White | 13 | 13 | 26 |
| Racial Category: Total of all subjects | 14 | 14 | 28 |

Ethnic Categories:

**Hispanic or Latino** – a person of Cuban, Mexican, Puerto Rican, South or Central American, or other Spanish culture or origin, regardless of race. The term "Spanish origin" can also be used in addition to "Hispanic or Latino."

#### **Not Hispanic or Latino**

Racial Categories:

**American Indian or Alaskan Native** – a person having origins in any of the original peoples of North, Central, or South America, and who maintains tribal affiliations or community attachment.

Asian – a person having origins in any of the original peoples of the Far East, Southeast Asia, or the Indian subcontinent including, for example, Cambodia, China, India, Japan, Korea, Malaysia, Pakistan, the Philippine Islands, Thailand, and Vietnam. (Note: Individuals from the Philippine Islands have been recorded as Pacific Islanders in previous data collection strategies.)

Black or African American – a person having origins in any of the black racial

groups of Africa. Terms such as "Haitian" or "Negro" can be used in addition to "Black or African American."

Native Hawaiian or other Pacific Islander – a person having origins in any of the original peoples of Hawaii, Guam, Samoa, or other Pacific Islands.

**White** – a person having origins in any of the original peoples of Europe, the Middle East, or North Africa.

## 17.0 Pathology Considerations/Tissue Biospecimens

17.1 Summary Table of Research Tissue Specimens to be Collected for this Protocol

| Research Study<br>(Section for more<br>information) | Specimen Purpose<br>(check all that apply) | Mandatory<br>or Optional | Type of<br>Tissue to<br>Collect | Block, Slides,<br>Core, etc.<br>(# of each to<br>submit) | Baseline,<br>prior to<br>Cycle 1<br>Day 1* | Process<br>at site?<br>(Yes or<br>No) | Temperature<br>Conditions for<br>Storage<br>/Shipping |
|---|---|---|---|---|---|---|---|
| Patient-derived tumor organoid culture and studies (Section 17.2 and 17.3) | <ul><li>☑ Correlative</li><li>☐ Eligibility Confirmation</li><li>☐ Banking</li><li>☐ Other (specify)</li></ul> | Mandatory | Fresh<br>Tissue | 3 cores | X | No | Cold ice pack |
| Immunohistochemistry (section 17.2 and 17.3) | <ul><li>☑ Correlative</li><li>☐ Eligibility Confirmation</li><li>☐ Banking</li><li>☐ Other (specify)</li></ul> | Mandatory | Formalin<br>Fixed<br>Paraffin<br>Embedded | 1 block from 4 <sup>th</sup> core collected at same time as fresh tissue cores | X | No | Ambient |

<sup>\*</sup>If baseline biopsy cannot be done (e.g., because not medically feasible or lack of lab capacity), and PI agrees, patient is still eligible.

#### 17.2 Correlative Tissue Collection

17.21 Tissue Kits will be provided for this protocol.

Interventional radiologist performing image-guided core biopsy of targeted tumor for research will contact personnel at the assigned laboratory at each Mayo Clinic site to obtain tissue kits.

## 17.23 Fresh Tissue

- 17.231 Three cores of fresh tumor tissue will be submitted after registration and prior to Cycle 1 Day 1 of treatment.
- 17.232 Fresh tissue must be labeled with the protocol number, study patient ID number, and the time and date of the biopsy.
- 17.233 Fresh tissue must be collected and shipped according to specific instructions provided in tissue kit and the table above.
- 17.234 Fresh tissue must be stored in tissue media in cold ice pack (~0°C)

#### 17.23 Paraffin Embedded Tissue

- 17.231 One block of BTC tumor tissue from research biopsy will be submitted after registration and prior to Cycle 1 Day 1 of treatment.
- 17.232 Paraffin embedded tissue must be labeled with the protocol number, study patient ID number, and the time and date of the biopsy.
- 17.233 Paraffin embedded tissue must be collected and shipped according to specific instructions provided in the table above.
- 17.234 Paraffin embedded tissue can be stored at ambient temperature.

#### 17.24 Shipping

- 17.241 Verify that ALL sections of the Tissue Specimen Submission Form (see Forms Packet), BAP Requisition Form (provided in kit), and specimen collection labels are completed and filled in correctly. Enter information from the Tissue Specimen Submission Form into the remote data entry system within 7 days after specimen collection (see Forms Packet).
- 17.242 Fresh tissue specimens collected in tissue media should be shipped overnight in cold ice pack (~0°C) to the laboratory of

## 17.25 Processing

- 17.251 Paraffin embedded tissue block
  DLMP or BAP/PRC Shared Resource will process the paraffin embedded tissue specimens according to routine protocols.
- 17.252 Fresh tissue cores

The laboratory of will process the fresh tissue specimens.

The fresh tissue specimens will be minced into  $\sim 0.5$  mm fragments in 1 mL resuspension media. They will be digested to single cells and plated with Matrigel and culture media.

## 17.3 Background and Methodology

## 17.31 Patient-derived tumor organoid

Preclinical tumor models are important tools to study cancer biology, develop novel therapeutics, and provide information for treatment decisions. However currently available tumor models such as cell lines, transgenic mice and patient-derived xenograft (PDX) model have inherent limitations that can adversely affect the translation of preclinical findings to the clinic. Patient-derived tumor organoid is a 3-D cell culture which enables the establishment of *ex vivo* tumor model from scant core-needle biopsy specimen in a timely manner. These tumor organoids recapitulate both phenotypes and genotypes of the donor tumor. (Vlachogiannis et al. 2018) The laboratory of at our institution has successfully established such tumor organoids from corebiopsy tumor specimens donated by patients with metastatic cholangiocarcinoma. The established tumor organoids were ready for drug screening and related molecular studies within 4-6 weeks of the biopsy. Though the concordance

between treatment effect in tumor organoids and the clinical benefit observed in the donor patients have been reported, the role of tumor organoids has not been prospectively evaluated in clinical trials of patients with advanced BTCs. Here, we aim to 1) determine if drug response from a parallel *ex vivo* trial using patient-derived tumor organoid correlates with clinical response to trifluridine/tipiracil plus irinotecan and 2) to evaluate the role of thymidine kinase 1 in predicting the clinical response to trifluridine/tipiracil plus irinotecan (Edahiro et al. 2018; Yoshino et al. 2018) and discover potential mechanisms of resistance and sensitivity.

MC1941 61 MCCC Amendment 1

#### 18.0 Records and Data Collection Procedures

#### 18.1 Submission Timetable

Data submission instructions for this study can be found in the Data Submission Schedule.

## 18.2 Event monitoring

See <u>Section 4</u> Test Schedule and Data Submission Schedule (DSS) for the event monitoring schedule.

## 18.3 CRF completion

This study will use Medidata Rave® for remote data capture (rdc) of all study data.

## 18.4 Site responsibilities

Each site will be responsible for insuring that <u>all materials</u> contain the patient's initials, MCCC registration number, and MCCC protocol number. Patient's name must be removed.

## 18.5 Supporting documentation

This study requires baseline supporting documentation of histologic diagnosis and staging of genetic mutations (genetic sequencing report), which includes the most recent tumor tissue biopsy pathology report. To submit these materials, they can be uploaded into the Supporting Documentation form in Medidata Rave®. These reports should be submitted within 21 days of registration.

This study requires supporting documentation for evidence of response to study therapy and progression after study therapy. Documentation of tumor genetic mutations is requested at any time, if available.

## 18.6 Labeling of materials

Each site will be responsible for insuring that <u>all materials</u> contain the patient's initials, MCCC registration number, and MCCC protocol number. Patient's name must be removed.

## 18.7 Incomplete materials

Any data entered into a form will result in that form being marked as "received." However, missing data in each form will be flagged by edit checks in the database.

## 18.8 Overdue lists

A list of overdue materials is automatically available to each site at any time. In addition, a list of overdue materials and forms for study patients will be generated monthly. The listings will be sorted by location and will include the patient study registration number. The appropriate co-sponsor/participant will be responsible to obtain the overdue material.

#### 18.9 Corrections forms

If a correction is necessary the QAS will query the site. The query will be sent to the appropriate site to make the correction in the database and respond back to the QAS.

MC1941 62 MCCC Amendment 1

## 19.0 Budget

19.1 Costs charged to patient: routine clinical care

Routine clinical care costs will be the responsibility of the patient and/or the patient's insurance company. This responsibility includes costs associated with surgery and with the administration of standard chemotherapy (such as irinotecan), and radiotherapy. These drugs are commercially available and will be the responsibility of the patient and/or the patient's insurance company.

#### 19.2 Tests to be research funded:

- Trifluridine/tipiracil will be provided by Taiho Oncology
- Research biopsy performed after registration and prior to treatment on Cycle 1, Day 1
- Correlative studies
- Collection, processing and storage of blood for research.

## 19.3 Other budget concerns:

Taiho Oncology will provide a grant through NCCN to Mayo Clinic to help with costs for the conduct of this study.

Mayo Clinic Cancer Center will provide Development funding to cover additional costs associated with the conduct of this study.

## 20.0 References

Bijnsdorp, Irene V.; Peters, Godefridus J.; Temmink, Olaf H.; Fukushima, Masakazu; Kruyt, Frank A. (2010): Differential activation of cell death and autophagy results in an increased cytotoxic potential for trifluorothymidine compared to 5-fluorouracil in colon cancer cells. In *International journal of cancer* 126 (10), pp. 2457–2468. DOI: 10.1002/ijc.24943.

Choi, C. W.; Choi, I. K.; Seo, J. H.; Kim, B. S.; Kim, J. S.; Kim, C. D. et al. (2000): Effects of 5-fluorouracil and leucovorin in the treatment of pancreatic-biliary tract adenocarcinomas. In *American journal of clinical oncology* 23 (4), pp. 425–428.

Dawson, Sarah-Jane; Tsui, Dana W. Y.; Murtaza, Muhammed; Biggs, Heather; Rueda, Oscar M.; Chin, Suet-Feung et al. (2013): Analysis of circulating tumor DNA to monitor metastatic breast cancer. In *The New England journal of medicine* 368 (13), pp. 1199–1209. DOI: 10.1056/NEJMoa1213261.

Diehl, Frank; Li, Meng; Dressman, Devin; He, Yiping; Shen, Dong; Szabo, Steve et al. (2005): Detection and quantification of mutations in the plasma of patients with colorectal tumors. In *Proceedings of the National Academy of Sciences of the United States of America* 102 (45), pp. 16368–16373. DOI: 10.1073/pnas.0507904102.

Diehl, Frank; Schmidt, Kerstin; Choti, Michael A.; Romans, Katharine; Goodman, Steven; Li, Meng et al. (2008): Circulating mutant DNA to assess tumor dynamics. In *Nature medicine* 14 (9), pp. 985–990. DOI: 10.1038/nm.1789.

Edahiro, Keitaro; Iimori, Makoto; Kobunai, Takashi; Morikawa-Ichinose, Tomomi; Miura, Daisuke; Kataoka, Yuki et al. (2018): Thymidine Kinase 1 Loss Confers Trifluridine Resistance without Affecting 5-Fluorouracil Metabolism and Cytotoxicity. In *Molecular cancer research : MCR* 16 (10), pp. 1483–1490. DOI: 10.1158/1541-7786.MCR-17-0686.

Emura, Tomohiro; Nakagawa, Fumio; Fujioka, Akio; Ohshimo, Hideyuki; Yokogawa, Tatsushi; Okabe, Hiroyuki; Kitazato, Kenji (2004a): An optimal dosing schedule for a novel combination antimetabolite, TAS-102, based on its intracellular metabolism and its incorporation into DNA. In *International journal of molecular medicine* 13 (2), pp. 249–255.

Emura, Tomohiro; Suzuki, Norihiko; Yamaguchi, Masahiro; Ohshimo, Hideyuki; Fukushima, Masakazu (2004b): A novel combination antimetabolite, TAS-102, exhibits antitumor activity in FU-resistant human cancer cells through a mechanism involving FTD incorporation in DNA. In *International journal of oncology* 25 (3), pp. 571–578.

Feisthammel, Jürgen; Schoppmeyer, Konrad; Mössner, Joachim; Schulze, Manfred; Caca, Karel; Wiedmann, Marcus (2007): Irinotecan with 5-FU/FA in advanced biliary tract adenocarcinomas: a multicenter phase II trial. In *American journal of clinical oncology* 30 (3), pp. 319–324. DOI: 10.1097/01.coc.0000258124.72884.7a.

Glimelius, B.; Hoffman, K.; Sjödén, P. O.; Jacobsson, G.; Sellström, H.; Enander, L. K. et al. (1996): Chemotherapy improves survival and quality of life in advanced pancreatic and biliary cancer. In *Annals of oncology : official journal of the European Society for Medical Oncology* 7 (6), pp. 593–600.

Guion-Dusserre, Jean-Florian; Lorgis, Veronique; Vincent, Julie; Bengrine, Leila; Ghiringhelli, Francois (2015): FOLFIRI plus bevacizumab as a second-line therapy for metastatic intrahepatic cholangiocarcinoma. In *World journal of gastroenterology* 21 (7), pp. 2096–2101. DOI: 10.3748/wjg.v21.i7.2096.

Hollebecque, Antoine; Calvo, Aitana; Andre, Thierry; Argiles, Guillem; Cervantes, Andres; Leger, Catherine et al. (2018): Phase I multicenter, open-label study to establish the maximum tolerated dose

(MTD) of trifluridine/tipiracil (TAS-102) and oxaliplatin combination in patients (pts) with metastatic colorectal cancer (mCRC). In *Journal of Clinical Oncology* 36 (4\\_suppl), p. 816. DOI: 10.1200/JCO.2018.36.4\ suppl.816.

Huggett, Matthew T.; Passant, Helen; Hurt, Chris; Pereira, Stephen P.; Bridgewater, John; Mukherjee, Somnath (2014): Outcome and patterns of care in advanced biliary tract carcinoma (ABC): experience from two tertiary institutions in the United Kingdom. In *Tumori* 100 (2), pp. 219–224. DOI: 10.1700/1491.16421.

Kim, Seung Tae; Lee, Won Suk; Lanman, Richard B.; Mortimer, Stefanie; Zill, Oliver A.; Kim, Kyoung-Mee et al. (2015): Prospective blinded study of somatic mutation detection in cell-free DNA utilizing a targeted 54-gene next generation sequencing panel in metastatic solid tumor patients. In *Oncotarget* 6 (37), pp. 40360–40369.

Larsen, Finn Ole; Markussen, Alice; Diness, Laura V.; Nielsen, Dorte (2018): Efficacy and Safety of Capecitabine, Irinotecan, Gemcitabine, and Bevacizumab as Second-Line Treatment in Advanced Biliary Tract Cancer: A Phase II Study. In *Oncology* 94 (1), pp. 19–24. DOI: 10.1159/000479970.

Lenz, Heinz-Josef; Stintzing, Sebastian; Loupakis, Fotios (2015): TAS-102, a novel antitumor agent: a review of the mechanism of action. In *Cancer treatment reviews* 41 (9), pp. 777–783. DOI: 10.1016/j.ctrv.2015.06.001.

Lesniewski-Kmak, K.; Moiseenko, V.; Saunders, M.; Wasan, H.; Argiles, G.; Borg, C. et al. (2018): O-022Phase II study evaluating trifluridine/tipiracil + bevacizumab and capecitabine + bevacizumab in first-line unresectable metastatic colorectal cancer (mCRC) patients who are non-eligible for intensive therapy (TASCO1): Results of the primary analysis. In *Annals of oncology : official journal of the European Society for Medical Oncology* 29 (suppl\_5). DOI: 10.1093/annonc/mdy149.021.

Liu, Minetta C. (2014): By the numbers: does circulating tumor cell enumeration have a role in metastatic breast cancer? In *Journal of clinical oncology : official journal of the American Society of Clinical Oncology* 32 (31), pp. 3479–3482. DOI: 10.1200/JCO.2014.56.6851.

Liu, Minetta C.; Shields, Peter G.; Warren, Robert D.; Cohen, Philip; Wilkinson, Mary; Ottaviano, Yvonne L. et al. (2009): Circulating tumor cells: a useful predictor of treatment efficacy in metastatic breast cancer. In *Journal of clinical oncology : official journal of the American Society of Clinical Oncology* 27 (31), pp. 5153–5159. DOI: 10.1200/JCO.2008.20.6664.

Mayer, Robert J.; van Cutsem, Eric; Falcone, Alfredo; Yoshino, Takayuki; Garcia-Carbonero, Rocio; Mizunuma, Nobuyuki et al. (2015): Randomized trial of TAS-102 for refractory metastatic colorectal cancer. In *The New England journal of medicine* 372 (20), pp. 1909–1919. DOI: 10.1056/NEJMoa1414325.

Murakami, Y.; Kazuno, H.; Emura, T.; Tsujimoto, H.; Suzuki, N.; Fukushima, M. (2000): Different mechanisms of acquired resistance to fluorinated pyrimidines in human colorectal cancer cells. In *International journal of oncology* 17 (2), pp. 277–283.

Rogers, Jane E.; Law, Lindsey; van Nguyen, D.; Qiao, Wei; Javle, Milind M.; Kaseb, Ahmed; Shroff, Rachna T. (2014): Second-line systemic treatment for advanced cholangiocarcinoma. In *Journal of gastrointestinal oncology* 5 (6), pp. 408–413. DOI: 10.3978/j.issn.2078-6891.2014.072.

Sanz-Altamira, P. M.; O'Reilly, E.; Stuart, K. E.; Raeburn, L.; Steger, C.; Kemeny, N. E.; Saltz, L. B. (2001): A phase II trial of irinotecan (CPT-11) for unresectable biliary tree carcinoma. In *Annals of oncology : official journal of the European Society for Medical Oncology* 12 (4), pp. 501–504.

Sharma, Atul; Dwary, Amit Dutt; Mohanti, Bidhu Kalyan; Deo, Surya V.; Pal, Sujoy; Sreenivas, Vishnu et al. (2010): Best supportive care compared with chemotherapy for unresectable gall bladder cancer: a

randomized controlled study. In *Journal of clinical oncology : official journal of the American Society of Clinical Oncology* 28 (30), pp. 4581–4586. DOI: 10.1200/JCO.2010.29.3605.

Shitara, Kohei; Doi, Toshihiko; Dvorkin, Mikhail; Mansoor, Wasat; Arkenau, Hendrik-Tobias; Prokharau, Aliaksandr et al. (2018): Trifluridine/tipiracil versus placebo in patients with heavily pretreated metastatic gastric cancer (TAGS): a randomised, double-blind, placebo-controlled, phase 3 trial. In *The Lancet. Oncology* 19 (11), pp. 1437–1448. DOI: 10.1016/S1470-2045(18)30739-3.

Siegel, Rebecca L.; Miller, Kimberly D.; Jemal, Ahmedin (2018): Cancer statistics, 2018. In *CA: a cancer journal for clinicians* 68 (1), pp. 7–30. DOI: 10.3322/caac.21442.

Tanaka, Nozomu; Sakamoto, Kazuki; Okabe, Hiroyuki; Fujioka, Akio; Yamamura, Keisuke; Nakagawa, Fumio et al. (2014): Repeated oral dosing of TAS-102 confers high trifluridine incorporation into DNA and sustained antitumor activity in mouse models. In *Oncology reports* 32 (6), pp. 2319–2326. DOI: 10.3892/or.2014.3487.

Ueno, H.; Okusaka, T.; Ikeda, M.; Takezako, Y.; Morizane, C. (2004): Phase II study of S-1 in patients with advanced biliary tract cancer. In *British journal of cancer* 91 (10), pp. 1769–1774. DOI: 10.1038/sj.bjc.6602208.

Valle, Juan; Wasan, Harpreet; Palmer, Daniel H.; Cunningham, David; Anthoney, Alan; Maraveyas, Anthony et al. (2010): Cisplatin plus gemcitabine versus gemcitabine for biliary tract cancer. In *The New England journal of medicine* 362 (14), pp. 1273–1281. DOI: 10.1056/NEJMoa0908721.

Varghese, Anna M.; Cardin, Dana B.; Hersch, Jon; Benson, Al B.; Hochster, Howard S.; Winkler, Robert et al. (2018a): Abstract CT062: A phase I dose escalation study of trifluridine and tipiracil (FTD/TPI) in combination with irinotecan (IRI) in patients with advanced gastrointestinal (GI) tumors. In *Cancer Res* 78 (13 Supplement), CT062-CT062. DOI: 10.1158/1538-7445.AM2018-CT062.

Varghese, Anna M.; Cardin, Dana Backlund; Hersch, Jonathan; Benson, Al Bowen; Hochster, Howard S.; Winkler, Robert E. et al. (2018b): A phase I expansion study of trifluridine and tipiracil (FTD/TPI) in combination with irinotecan (IRI) and bevacizumab (BEV) in patients with metastatic colorectal cancer (mCRC). In *Journal of Clinical Oncology* 36 (15\\_suppl), p. 3546. DOI: 10.1200/JCO.2018.36.15\ suppl.3546.

Vlachogiannis, Georgios; Hedayat, Somaieh; Vatsiou, Alexandra; Jamin, Yann; Fernández-Mateos, Javier; Khan, Khurum et al. (2018): Patient-derived organoids model treatment response of metastatic gastrointestinal cancers. In *Science* 359 (6378), pp. 920–926. DOI: 10.1126/science.aao2774.

Yoshino, Takayuki; Yamazaki, Kentaro; Shinozaki, Eiji; Komatsu, Yoshito; Nishina, Tomohiro; Baba, Hideo et al. (2018): Relationship Between Thymidine Kinase 1 Expression and Trifluridine/Tipiracil Therapy in Refractory Metastatic Colorectal Cancer: A Pooled Analysis of 2 Randomized Clinical Trials. In *Clinical colorectal cancer* 17 (4), e719-e732. DOI: 10.1016/j.clcc.2018.07.009.

Zheng, Yi; Tu, Xiaoxuan; Zhao, Peng; Jiang, Weiqin; Liu, Lulu; Tong, Zhou et al. (2018): A randomised phase II study of second-line XELIRI regimen versus irinotecan monotherapy in advanced biliary tract cancer patients progressed on gemcitabine and cisplatin. In *British journal of cancer* 119 (3), pp. 291–295. DOI: 10.1038/s41416-018-0138-2.

MC1941 66 MCCC Amendment 1

## **Appendix I ECOG Performance Status**

| ECOG PERFORMANCE STATUS* | |
|---|---|
| Grade | ECOG |
| 0 | Fully active, able to carry on all pre-disease performance without restriction |
| 1 | Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work |
| 2 | Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours |
| 3 | Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours. |
| 4 | Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair. |
| 5 | Dead |

<sup>\*</sup>As published in Am. J. Clin. Oncol.:

Oken, M.M., Creech, R.H., Tormey, D.C., Horton, J., Davis, T.E., McFadden, E.T., Carbone, P.P.: Toxicity And Response Criteria Of The Eastern Cooperative Oncology Group. Am J Clin Oncol 5:649-655, 1982.

The ECOG Performance Status is in the public domain therefore available for public use. To duplicate the scale, please cite the reference above and credit the

| _ |
|----------|
| From |
| From |
| 1 1 0111 |

# Appendix II Patient Medication Diary

| <b>Name</b> | | | | | | Sti | idy ID | Numbe | er | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Please con<br>took in the | - | | • | • | sis. Wri | te in the | amoun | t of the | dose of | f TAS-1 | 02 that | you |
| On the day<br>daily dose<br>scheduled | , please | | | • | • | - | | | - | _ | • | |
| If you exp<br>please reco | | • | | dical co | mplaint | ts or tak | e any m | edicatio | on other | than T | AS-102 | |
| Cycle | | | | | | | | | | | | |
| Week of: | | | | | _ | | | | | | | |
| TAS-102 | Da | y 1 | Da | y 2 | Da | ıy 3 | Da | y 4 | Da | y 5 | Day<br>6 | Day 7 |
| FTD-TPI | AM | PM | AM | PM | AM | PM | AM | PM | AM | PM | | |
| 15mg<br>tablets | | | | | | | | | | | | |
| 20mg<br>tablets | | | | | | | | | | | | |
| | | | | | <u> </u> | | | | | | | |
| Week of: | | | | | _ | | | | | | | |
| TAS-102 | Da | ıy 8 | Day 9 | Da | ıy 10 | Day 1 | 1 D | ay 12 | Day 1 | 13 D | ay 14 | ] |
| FTD-TPI | | | | | | | | | | | | |
| Patient signature: | | | | | | | | | | | | |
| | M | y next s | schedul | ed visit | is: | | | | | | | |
| | If | you ha | ve any q | uestion | s, pleas | se call: _ | | | | | | |
| Nambar - f | milla ==4 | | | | | linator U | | | | | | |
| Number of Discrepanc | - | urned<br>/No_ | | | umber of<br>Terified b | of vials re | aumed: | | –<br>Dat | te | | |